

Title: Lotriga Granular Capsules Special Drug Use Surveillance [Long-term use survey]

NCT Number: NCT02153073

Statistical analysis plan Approve Date: 22-Sep-2017

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

## Statistical Analysis Plan

## (for Periodic Safety Reporting/Reexamination Application)

<Lotriga Granular Capsules>

[Long-term use]

Takeda Pharmaceutical Company Limited Japan Development Center Director of Biostatistics Division



Ver. 4.0: Prepared on September 22, 2017

#### Table of Contents

| 1.0 | Defini | tions of Terms | 1 |
|---|---|---|---|
| 1.1 | Def | initions | 1 |
| 1.2 | Nur | nber of Display Digits | 5 |
| 1.3 | Con | fidence Coefficient. | 5 |
| 1.4 | Har | ndling of Evaluation Timepoint Data | 6 |
| 2.0 | Resul | ts of Special Drug Use Surveillance (Survey 1) | 7 |
| 2.1 | Pat | ient Breakdown (Patient Disposition) | 7 |
| 2.2 | Pat | ient Demographics | 8 |
| 2.3 | Trea | atment Details | 0 |
| 2.4 | Safe | ety Statistical Analysis1 | 2 |
| 2 | 2.4.1 | Onset Status of Adverse Drug Reactions or Infections (Exhibit 2) | 2 |
| 2 | 2.4.2 | Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients 1 | 4 |
| 2 | 2.4.3 | Onset Status of AE | 4 |
| 2 | 2.4.4 | Onset Status of Adverse Events in Safety-Unevaluable Patients | 5 |
| 2 | 2.4.5 | Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, an | d |
| ( | Outcom | e1 | 5 |
| 2 | 2.4.6 | Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome | 6 |
| 2 | 2.4.7 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness | 3, |
| ( | Onset T | ime, and Outcome1 | 6 |
| 2 | 2.4.8 | Rate of Patients of Adverse Drug Reactions or Infections by Patient Demographics an | d |
| 7 | [reatme | ent Details1 | 7 |
| 2 | 2.4.9 | Onset Status of Adverse Drug Reactions or Infections by Sex Group 1 | 8 |
| 2 | 2.4.10 | Onset Status of Adverse Drug Reactions or Infections by Age Group | 9 |
| 2 | 2.4.11 | Onset Status of Adverse Drug Reactions or Infections by BMI | 9 |
| 2 | 2.4.12 | Onset Status of Adverse Drug Reactions or Infections by Complications | 9 |
| 2 | 2.4.13 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of | f |
| I | Hyperte | nsion Complications1 | 9 |
| 2 | 2.4.14 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of | f |
| I | Diabete | s Complications | 0 |
| 2 | 2.4.15 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Live | r |
| ( | Complic | ations2 | 0 |
| 2 | 2.4.16 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of | f |
| I | Kidney | Complications | 0 |
| 2 | 2.4.17 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of | f |
| ( | Cardiac | Complications | 0 |
| 2 | 2.4.18 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of | f |
| ( | Cerebro | vascular Complications | 1 |

| 2.4.19 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
|---|---|
| Bleedin | g-related Event Complications |
| 2.4.20 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Anticoagulant and/or Antiplatelet Drugs |
| 2.4.21 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or |
| Absence | e of Concomitant Anticoagulant and/or Antiplatelet Drugs |
| 2.4.22 | Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride |
| Level | 23 |
| 2.4.23 | Onset Status of Adverse Drug Reactions or Infections by Baseline Random |
| Triglyce | ride Level |
| 2.4.24 | Onset Status of Adverse Drug Reactions or Infections by Initial Dose |
| 2.4.25 | Onset Status of Adverse Drug Reactions or Infections by Breakdown of Change in |
| Daily D | ose |
| 2.4.26 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Antihyperlipidemic Drug Use (during observation period)24 |
| 2.4.27 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Statins Drugs |
| 2.4.28 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Fibrate Drugs24 |
| 2.4.29 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Intestinal Transporter Inhibitors |
| 2.4.30 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Anion-exchange Resin |
| 2.4.31 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Nicotinic Acid Derivatives |
| 2.4.32 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Probucol |
| 2.4.33 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of |
| Concom | itant Ethyl Icosapentate (EPA) |
| 2.4.34 | Changes in Laboratory Test Values (Glucose Metabolism) |
| 2.4.35 | Changes in Laboratory Test Values (Glucose Metabolism) <with diabetic<="" td=""></with> |
| Complic | eations> |
| 2.4.36 | Changes in Laboratory Test Values (Glucose Metabolism) <without diabetic<="" td=""></without> |
| Complic | eations> |
| 2.4.37 | Summary of Onset Status of Serious Adverse Events (Exhibit 2-2) |
| 2.4.38 | Summary of Onset Status of Serious Adverse Drug Reactions or Infections |
| 2.4.39 | Summary of Onset Status of Serious Adverse Events in Safety-Unevaluable patients |
| | 30 |
| 2.4.40 | Summary of Onset Status of Serious Adverse Drug Reactions or Infections in |

| Safety- | Unevaluable patients |
|---|---|
| 2.5 Eff | icacy Statistical Analysis |
| 2.5.1 | Changes in Laboratory Test Values (Fasting Lipid) |
| 2.5.2 | Changes in Laboratory Test Values (Random Lipid) |
| 2.5.3 | Changes in Laboratory Test Values (Lipid) |
| 2.5.4 | Changes in Fasting Lipid-Related Ratio |
| 2.5.5 | Changes in Fasting Triglyceride by Patient Demographics and Treatment Details 34 |
| 2.5.6 | Changes in Random Triglyceride by Patient Demographics and Treatment Details 35 |

#### 1.0 Definitions of Terms

## 1.1 Definitions

| Item | Definition |
|---|---|
| Survey unit period | Periodic Safety Report 1: July 22, 2012 to January 21, 2013 |
| (periodic safety report) | Periodic Safety Report 2: January 22, 2013 to July 21, 2013 |
| | Periodic Safety Report 3: July 22, 2013 to January 21, 2014 |
| | Periodic Safety Report 4: January 22, 2014 to July 21, 2014 |
| | Periodic Safety Report 5: July 22, 2014 to July 21, 2015 |
| | Periodic Safety Report 6: July 22, 2015 to July 21, 2016 |
| | Periodic Safety Report 7: July 22, 2016 to July 21, 2017 |
| | Periodic Safety Report 8: July 22, 2017 to July 21, 2018 |
| Drug | Lotriga Granular Capsules |
| SOC | System organ class of MedDRA. |
| HLGT | High level group term of MedDRA. |
| PT | Preferred term of MedDRA. |
| LLT | Lowest level term of MedDRA. |
| Enrolled patient | A patient approved for enrollment in the Study. |
| Patient with eCRF | An enrolled patient whose eCRF was submitted via |
| collected | |
| Patient with eCRF | An enrolled patient other than a patient with eCRF collected. |
| uncollected | |
| Locked patient | A patient who has completed the approval process in the PMS system. |
| Unlocked patient | A patient with eCRF collected other than a locked patient. |
| Safety-evaluable patient | A locked patient included in safety evaluation. |
| Safety-unevaluable patient | A locked patient excluded from safety evaluation. |
| Efficacy-evaluable patient | A safety-evaluable patient included in efficacy evaluation. |
| Efficacy-unevaluable | A safety-evaluable patient excluded from efficacy evaluation. |
| patient | |
| ADR | An abbreviated form of the term 'adverse drug reaction or infection.' |
| | Refers to an adverse event other than those judged by the investigator as 'not |
| | related' in causality to the Drug. |
| | In this plan, 'adverse drug reactions or infections' is used in headings, and |
| | 'ADRs' is used in the text and tables. |
| Serious adverse event | [Prior-approval data] |
| (SAE) | An adverse event (AE) judged as 'serious' by the trial investigator. |
| | [Surveillance data] |
| | An adverse event (AE) judged as 'serious' by the investigator. |
| | Note that events listed in the separate MedDRA code list of the Takeda |
| | Medically Significant AE List should be treated as serious even if judged as |

| Item | Definition |
|---|---|
| | 'not serious' by the investigator. |
| Bleeding-related event | An event falling under Standardized MedDRA Query (SMQ) code 20000038 |
| | (hemorrhagic SMQ [narrow scope]). |
| Rate of patients | [For safety compilation with safety-evaluable patients] |
| | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Evaluable Patients] × 100. |
| | [For safety compilation with safety-unevaluable patients] |
| | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Unevaluable Patients] × 100. |
| Onset time | Calculated by the following equation: [Onset Date] - [Start Date] + 1. |
| | If the onset date is unknown, use the first day of the month as the onset date in |
| | this equation. However, use the start date as the onset date if [Start Year & |
| | Month] = [Onset Year & Month]. |
| Liver patient | A patient with 'fatty liver,' 'alcoholic fatty liver,' 'chronic hepatitis' or 'hepatic |
| | cirrhosis' check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SMQ code 20000005 (hepatic SMQ [narrow |
| | scope]) in the Complication Details (Other Diseases) field. |
| Kidney patient | A patient with 'diabetic nephropathy,' 'glomerulonephritis' or 'chronic kidney |
| | disease (CKD)' check-marked in the Complication Details field. Or a patient |
| | with a complication falling under the Takeda MedDRA query (TMQ) (Renal |
| | Disease) in the Complication Details (Other Diseases) field. |
| Heart patient | A patient with 'myocardial infarction,' 'angina pectoris' or 'atrial fibrillation' |
| | check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SOC code 10007541 (cardiac disorders) in the |
| | Complication Details (Other Diseases) field. |
| Cerebrovascular patient | A patient with 'cerebral infarction' or 'cerebral hemorrhage' check-marked in |
| | the Complication Details field. Or a patient with a complication falling under |
| | the SMQ code 20000060 (cerebrovascular SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Diabetic patient | A patient with 'diabetes' check-marked in the Complication Details field. Or a |
| | patient with a complication falling under the TMQ code (Diabetes Mellitus |
| | Confirmed diagnosis, excl diagnostics) in the Complication Details (Other |
| | Diseases) field. |
| Hypertensive patient | A patient with 'hypertension' check-marked in the Complication Details field. |
| | Or a patient with a complication falling under the SMQ code 20000147 |
| | (hypertensive SMQ [narrow scope]) in the Complication Details (Other |
| | Diseases) field. |
| Myocardial infarction | A patient with 'myocardial infarction' check-marked in the Complication |

| Item | Definition |
|---|---|
| patient | Details field. Or a patient with a complication falling under the SMQ code |
| | 20000047 (myocardial infarction SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Anginal patient | A patient with 'angina pectoris' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10002383 (angina pectoris), 10002388 (unstable angina pectoris), 10036759 |
| | (Prinzmetal angina), or 10058144 (postinfarction angina) in the Complication |
| | Details (Other Diseases) field. |
| Atrial fibrillation patient | A patient with 'atrial fibrillation' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10003658 (atrial fibrillation) in the Complication Details (Other Diseases) |
| | field. |
| Ischemic cerebrovascular | A patient with 'cerebral infarction' check-marked in the Complication Details |
| patient | field. Or a patient with a complication falling under the SMQ code 20000063 |
| | (ischemic cerebrovascular disease SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Hemorrhagic | A patient with 'cerebral hemorrhage' check-marked in the Complication Details |
| cerebrovascular patient | field. Or a patient with a complication falling under the SMQ code 20000064 |
| | (hemorrhagic cerebrovascular disease SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Bleeding-related event | A patient with a complication falling under the SMQ code 20000038 (bleeding |
| patient | SMQ [narrow scope]) in the Complication Details (Other Diseases) field. |
| Age | Calculated by the following equation: [Start Year] - [Birth Year] - 1 if [Start |
| | Month & Day] < [Birth Month & Day]. |
| | Calculated by the following equation: [Start Year] - [Birth Year] if [Start Month |
| | & Day] ≥ [Birth Month & Day]. |
| | If the birth day is unknown, use the first day of the month instead in this |
| | equation. |
| BMI | Calculated by the following equation: [Weight (kg)] / (0.0001 × [Height (cm)] |
| | × [Height (cm)]). Indicated by rounding off to the first decimal place. |
| Disease duration (in years) | Calculated by the following equation: ([Start Year & Month] - [Year & Month] |
| | of Hyperlipidemia Diagnosis] + 1) / 12. Indicated by rounding off to the first |
| | decimal place. |
| Start date | The start date of first administration of the Drug stated in the Treatment |
| | Duration field of the eCRF. |
| End date | The end date of last administration of the Drug stated in the Treatment Duration |
| | field of the eCRF. |
| | However, if the end date of last administration is in 'ongoing 12 months after |

| Item | Definition |
|---|---|
| | baseline,' the end date should be the start date plus 405 days. |
| Observation period (in | Refers to the entire period of observation. The start date and end date of |
| days) | observation period should be the same as the 'start date' and 'end date,' |
| | respectively. |
| | Calculated by the following equation: [End Date] - [Start Date] + 1. |
| Treatment duration (in | Refers to the entire period of treatment. A total of Drug dosing periods in the |
| days) | number of actual administration days, excluding washout period. Calculated as |
| | a total of ([End Date] - [Start Date] + 1) in the number of actual administration |
| | days, excluding washout period. |
| Mean daily dose | Calculated by the following equation: Total of ([Daily Dose] × [Total Period of |
| | Treatment with the Dose]) / [Observation Period]. See the above for calculation |
| | of observation period. |
| Concomitant medication | A drug used during the surveillance period. However, concomitant medications |
| | exclude drugs used for adverse events occurring during the period. |
| Antihyperlipidemic drug | A drug starting with any of the following drug codes: 218, 2190006, 2190101, |
| | 2190102, 2190103, 2190104, 290006, 3133001, 3133400, 3399004. |
| Statins drug | A drug starting with any of the following drug codes: 2189010, 2189011, |
| | 2189012, 2189015, 2189016, 2189017. |
| Fibrate drug | A drug starting with drug code: 2183. |
| Intestinal transporter | A drug starting with drug code: 2189018. |
| inhibitor | |
| Anion-exchange resin | A drug starting with any of the following drug codes: 2189009, 2189014. |
| Nicotinic acid derivative | A drug starting with any of the following drug codes: 2189004, 2189005, |
| | 2190006. |
| Probucol | A drug starting with drug code: 2189008. |
| Ethyl icosapentate (EPA) | A drug starting with drug code: 3399004. |
| Anticoagulant drug | A drug starting with any of the following drug codes: 333, 2190408, 6343424. |
| Antiplatelet drug | A drug starting with any of the following drug codes: 3399 (excluding |
| | 3399004), 2171010, 2171402. |
| Anticoagulant/antiplatelet | A drug that falls under the class of either anticoagulant or antiplatelet drugs |
| drug | |
| LDL cholesterol | Calculated the equation below if the patient is fasting at the time of blood |
| (Friedewald formula) | collection for laboratory testing with triglyceride 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol - triglyceride / 5 |
| Non-HDL cholesterol | Calculated by the equation below if triglyceride is 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol |

| Item | Definition |
|---|---|
| TC/HDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | Total cholesterol / HDL cholesterol |
| LDL-C/HDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / HDL cholesterol |
| LDL-C/Apo-B ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / Apo-B (fasting) |
| Summary statistics | Number of patients, mean value, standard deviation, minimum value, first |
| | quartile, median, third quartile, maximum value |

#### 1.2 Number of Display Digits

| Item | Definition |
|---|---|
| Percentage (%) | Rate of patients with ADRs: |
| | Indicated by rounding off to the second decimal place. |
| | Other than above: |
| | Indicated by rounding off to the first decimal place. |
| Summary statistics Mean value: | |
| | Indicated by rounding off to the first digit below the raw numerical data. |
| | Standard deviation: |
| | Indicated by rounding off to the second digit below the raw numerical data. |
| | First quartile, median, third quartile: |
| | Indicated by rounding off to the first digit below the raw numerical data. |
| | Minimum value, maximum value: |
| | Indicated at the same digits of the raw numerical data. |
| Confidence interval | Indicated by rounding off to the second digit below the raw numerical data. |

#### 1.3 Confidence Coefficient

Two-sided 95%

#### 1.4 Handling of Evaluation Timepoint Data

The evaluation timepoints are the start of treatment with the Drug (baseline), Month 3, Month 6, Month 9, Month 12, and final evaluation timepoint.

If multiple data exist within each evaluation timepoint, calculate absolute values of difference in measurement intervals from the basic day count and adopt the minimum absolute value as date for that evaluation timepoint. If all the absolute values are the same, adopt one for the latest date of testing/measurement. Test/Measurement values should not be adopted that have been obtained after completion of treatment with the Drug. The final evaluation timepoint test/measurement should be one taken on the latest date within 405 days elapsed since the start date (including values tested/measured during washout period). Note that the number days elapsed since the start date should be counted with the start date as day 0 and the previous day as day -1.

| Evaluation Timepoint | Tolerance (Number of Days Since Baseline) | Basic Day Count |
|---|---|---|
| Baseline | -90 to 0 | 0 |
| Month 3 | 1 to 135 | 90 |
| Month 6 | 136 to 225 | 180 |
| Month 9 | 226 to 315 | 270 |
| Month 12 | 316 to 405 | 360 |
| Final evaluation | 1 to 405 | - |
| timepoint | | |

#### 2.0 Results of Special Drug Use Surveillance (Survey 1)

<Lotriga Granular Capsules Special Drug Use Surveillance [long-term use survey]>

### 2.1 Patient Breakdown (Patient Disposition)

| Statistical Analysis | Enrolled patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Number of enrolled patients, number of patient enrollment sites, number of patients |
| Statistical Analysis | with eCRFs collected, number of patients with eCRFs uncollected, number of locked |
| | patients, number of unlocked patients, number of safety-evaluable patients, number of |
| | safety-unevaluable patients, number of efficacy-evaluable patients, number of |
| | efficacy-unevaluable patients |
| | Do not double-count the same medical institution with different participating clinical |
| | departments when counting the number of patient enrollment sites. |
| | Count the number of patients per reason below for not collecting and total the |
| | numbers when the number of patients with eCRFs uncollected. |
| | <reasons collecting="" for="" not=""></reasons> |
| | Survey under way |
| | eCRFs uncollectable |
| | Investigator transferred |
| | • Investigator's health reasons |
| | Patients enrolled 15 days after Drug prescription [before eCRF collection] |
| | • Others |
| | Count the number of patients per reason below for exclusion and total the numbers |
| | when counting the numbers of safety- and efficacy-unevaluable patients. If the same |
| | patient falls under multiple reasons for exclusion, they should be counted separately. |
| | <reasons evaluation="" exclusion="" for="" from="" safety=""></reasons> |
| | Drug administered before contract period |
| | Patient enrolled 15 days after Drug prescription |
| | No data available after Drug administration |
| | • Drug not administered |
| | <reasons efficacy="" evaluation="" exclusion="" for="" from=""></reasons> |
| | Other than target disease |
| | • Exclusion criteria violation |
| | No output needs to be generated for items for which the number of patients is zero. |
| | For periodic safety reports, the numbers of efficacy-evaluable and unevaluable |
| D' (D 11 ) | patients should not be counted. |
| Figure/Table No. | Figure 2.1, Table 2.1 |

### 2.2 Patient Demographics

| Statistical Analysis | Safaty avaluable nationts | in this enacial drug use surveillance |
|---|---|---|
| Set Statistical Allarysis | Safety-evaluable patients in this special drug use surveillance | |
| Details of | Categorize the patient population by the following categories for each item and | |
| Statistical Analysis | | |
| Statistical / Marysis | compile the number of patients and incidence. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Summary statistics |
| | | Minimum age to 64 years, 65 to 74 years, 75 years to |
| | | maximum age, Unknown |
| | Treatment category | Outpatient, inpatient |
| | BMI | Summary statistics |
| | | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to |
| | | less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | | Hypertension, Diabetic, Liver disorder, Kidney |
| | | disorder, Cardiac disorders [myocardial infarction, |
| | Complication | angina pectoris, atrial fibrillation, others], |
| | breakdown | Cerebrovascular diseases [hemorrhagic |
| | | cerebrovascular disease, ischemic cerebrovascular |
| | | disease, others], Bleeding-related event, Others |
| | Drinking history | |
| | (Does the patient | |
| | drink alcoholic | Yes, No, Unknown |
| | beverages nearly | |
| | every day?) | |
| | Fasting triglyceride at | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured |
| | baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured |

| | | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
|---|---|---|
| | Smoking history | Never, Current, Former, Unknown |
| | Hypersensitivity disposition | No, Yes, Unknown |
| | | Summary statistics |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence of surgery within one month before baseline | No, Yes |
| | Pregnancy status<br>during treatment (only<br>for female) | No, Yes |
| Figure/Table No. | Table 2.2 | <u>, </u> |

#### 2.3 Treatment Details

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set Details of Statistical Analysis | Categorize the patient population by the following categories for each item and compile the number of patients and incidence. | |
| | Item Name | Category |
| | Initial dose | 2 g, 4 g, Other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |
| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | Statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others |
| | Presence or absence of concomitant anticoagulant/antiplatelet drug use (during observation period) | No, Yes |
| | Breakdown of concomitant anticoagulant/antiplatelet drugs (during observation period) | Anticoagulant drugs, antiplatelet drugs |
| | Completion of treatment with the Drug | No, Yes |
| | Reason for treatment | Treatment goal achieved, AE developing, Patient no |

| | completion | longer visiting hospital due to hospital transfer or otherwise, Insufficient effect, Other |
|---|---|---|
| | | otherwise, insufficient effect, other |
| Figure/Table No. | Table 2.3 | |

## 2.4 Safety Statistical Analysis

### 2.4.1 Onset Status of Adverse Drug Reactions or Infections (Exhibit 2)

| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in | |
|---|---|---|
| Set | clinical studies in Japan used for safety evaluation stated in the Adverse Drug | |
| | Reactions section of the package insert) and this special drug use surveillance | |
| Details of | Compile the following items for the prior-approval status and per survey unit period | |
| Statistical Analysis | of the special drug use survei | llance. |
| | | er of study sites,' 'number of surveyed patients,' 'number |
| | - | 'number of ADRs' should cover safety-evaluable patients |
| | locked during each survey un | • |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients with ADRs | Number of patients in which ADRs occurred. |
| | N. 1. Gipp | Number of ADRs that occurred. |
| | Number of ADRs | Every PT occurring should be counted as one event. |
| | Data of nationts with | Calculated by the following equation: [Number of |
| | Rate of patients with ADRs | Patients with ADRs] / [Number of |
| | | Safety-Evaluable Patients] × 100 The calculation method in performing each |
| | | analysis should be as follows: |
| | | [Number of patients with ADRs] |
| | | • Number of patients in which ADRs occurred. [Number of ADRs] |
| | | • Number of ADRs that occurred. If the same ADR |
| | | occurs more than once in the same patient, a total of frequencies of the ADR should be counted. |
| | | [Rate of patients with ADRs] |
| | | • Calculated by the following equation: [Number of Patients with ADRs] / [Number of |
| | | Safety-Evaluable Patients] × 100. |
| | ADR type | [ADR type] |
| | J. J | • ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in |
| | | each category. If SOC is 'Investigations,' classify |
| | | by HLGT (sort by HLGT code in ascending order |
| | | but without outputting) and compile ADRs by PT. |
| | | • At SOC level, the numbers and rates of patients |
| | | with ADRs should be presented by SOC |
| | | internationally agreed order. If the same SOC |
| | | occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. |
| | | At PT level, the numbers and rates of patients with |
| | | ADRs should be presented by PT code in |

| | Cumulative total for special drug use surveillance | ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the PT. A respective total of the numbers of study sites and patients per survey unit period. Do not double-count the same medical institution when counting the number of study sites. |
|---|---|---|
| Figure/Table No. | Table 2.4.1 | |

#### 2.4.2 Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients

| Details of Statistical Analysis Tem Name Details of Statistical Analysis | Statistical Analysis | Safety-unevaluable patients in this specified drug use surveillance | |
|---|---|---|---|
| Statistical Analysis Number of study sites Number of medical institutions that have collected eCRFs | Set | | |
| Number of study sites Number of surveyed patients Number of patients with ADRs Number of patients with ADRs Number of ADRs Number of ADRs that have occurred. Number of ADRs that have occurred. Number of ADRs that have occurred. Every PT occurring should be counted as one event. The calculation method in performing each analysis should be as follows: [Number of ADRs] Number of ADRs] Number of ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [ADR type] ADR should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the PT. | Details of | Compile the following items. | |
| Number of study sites Number of surveyed patients Number of patients with ADRs Number of ADRs hat have occurred. Number of ADRs bounded as one event. The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] Number of ADRs bumber of patients in which ADRs occurred. [Number of patients with ADRs] Number of ADRs] Number of ADRs cocurred. [Number of ADRs] Number of ADRs bould be counted. [Number of ADRs] Number of ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. | Statistical Analysis | Item Name | Details of Statistical Analysis |
| Number of patients with ADRs Number of patients with ADRs that have occurred. Number of ADRs Description of ADRs that have occurred. Number of ADRs that have occurred. Every PT occurring should be counted as one event. The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] Number of patients in which ADRs occurred. [Number of ADRs] Number of ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [ADR type] ADR should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the PT. | | Number of study sites | |
| Number of ADRs that have occurred. Every PT occurring should be counted as one event. The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] • Number of patients in which ADRs occurred. [Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [ADR type] • ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient, ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient, ADRs should be counted as one patient, ADRs should be counted as one patient, ADRs should be counted as one patient in the PT. | | | Number of safety-unevaluable patients. |
| Number of ADRs Every PT occurring should be counted as one event. The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] Number of patients in which ADRs occurred. [Number of ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [ADR type] ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient, ADRs should be counted as one patient in the PT. | | I I | Number of patients in which ADRs occurred. |
| analysis should be as follows: [Number of patients with ADRs] Number of patients in which ADRs occurred. [Number of ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [ADR type] ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient, ADRs should be counted as one patient, ADRs should be counted as one patient, ADRs should be counted as one patient in the PT. | | Number of ADRs | Every PT occurring should be counted as one |
| Figure/Table No. Table 2.4.2 | | ADR type | The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] • Number of patients in which ADRs occurred. [Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [ADR type] • ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient, ADRs should be counted as one patient, ADRs should be counted as one patient in |
| O | Figure/Table No. | Table 2.4.2 | |

#### 2.4.3 Onset Status of AE

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | The compilation method is the same as described in section 2.4.1. However, adverse |
| Statistical Analysis | drug reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.3 |

#### 2.4.4 Onset Status of Adverse Events in Safety-Unevaluable Patients

| Statistical Analysis | Safety-unevaluable patients in this specified drug use surveillance |
|---|---|
| Set | |
| Details of | Compilation method is the same as described in section 2.4.2. However, adverse drug |
| Statistical Analysis | reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.4 |

### 2.4.5 Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize AD | Categorize ADRs by the following categories for each item and compile ADR types. |
| Statistical Analysis | Item Name Details of Statistical Analysis | |
| | Number of patients | Compile the number of patients with ADRs. |
| | Number of ADRs hould be compiled by totaling associated PTs that occurred. At PT level, every PT occurring should be counted as one event. | |
| | Item Name Category | |
| | Seriousness | Serious, Not serious |
| | Onset time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over, Unknown |
| | Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, Death, Unknown |
| Figure/Table No. | Table 2.4.5 | |

### 2.4.6 Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize AEs | by the following categories for each item and compile AE types. |
| Statistical Analysis | The compilation | on method of AE types is the same as described in section 2.4.5. |
| | However, adver | rse drug reactions should be replaced by adverse events. |
| | Item Name | Category |
| | Seriousness | Serious, Not serious |
| | Ongot time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to |
| | Onset time | 360 days, 361 days or over, Unknown |
| | Outcomo | Resolved, Resolving, Not resolved, Resolved with sequelae, |
| | Outcome Death, Unknown | |
| | Causal | Related, Not related, Unevaluable |
| | relationship | If AEs (LLTs) occur more than once in the same patient, they |
| | with the | should be counted as one event in the following order of priority: |
| | Drug | (1) Related, (2) Unevaluable, (3) Not related |
| Figure/Table No. | Table 2.4.6 | |

### 2.4.7 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Time,

#### and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Categorize adverse drug reactions (bleeding-related events) by the following |
| Statistical Analysis | categories for each item, and count the types of adverse drug reactions |
| | (bleeding-related events). |
| | The categories and the compilation method of adverse drug reactions are the same as |
| | described in section 2.4.5. |
| Figure/Table No. | Table 2.4.7 |

# 2.4.8 Rate of Patients of Adverse Drug Reactions or Infections by Patient Demographics and TreatmentDetails

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADRs by the following categories for each item and compile the rate of | |
| Statistical Analysis | patients with ADRs. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | ВМІ | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | Complication breakdown | Hypertension, Diabetic, Liver disorder, Kidney disorder, Cardiac disorders Cerebrovascular diseases, Bleeding-related event, Others |
| | Fasting triglyceride at | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured |
| | baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, |
| | | 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Initial dose | 2 g, 4 g, other |
| | Breakdown of presence of change in daily dose | |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |

| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), |
|---|---|---|
| | Presence or absence of concomitant anticoagulant/antiplatelet drug use (during observation period) | No, Yes |
| | Breakdown of concomitant anticoagulant/antiplatelet drugs (during observation period) | Anticoagulant drugs, antiplatelet drugs |
| Figure/Table No. | Table 2.4.8 | |

## 2.4.9 Onset Status of Adverse Drug Reactions or Infections by Sex Group

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Classify the patient population into males and females, and compile ADR types. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.9 |

#### 2.4.10Onset Status of Adverse Drug Reactions or Infections by Age Group

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Classify the patient population into 64 years or below, 65 to 74 years, and 75 years or |
| Statistical Analysis | over, and compile ADR types. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.10 |

#### 2.4.11 Onset Status of Adverse Drug Reactions or Infections by BMI

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Classify the patient population into less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , |
| Statistical Analysis | 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, and compile ADR types. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.11 |

#### 2.4.12 Onset Status of Adverse Drug Reactions or Infections by Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.12 |

#### 2.4.13 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Hypertension

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of hypertension complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.13 |

#### 2.4.14 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Diabetes

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of diabetes complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.14 |

#### 2.4.15 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Liver

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of liver complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.15 |

#### 2.4.16 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kidney

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of kidney complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.16 |

#### 2.4.17 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Cardiac

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of cardiac complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.17 |

# 2.4.18 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of CerebrovascularComplications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of cerebrovascular complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.18 |

# 2.4.19 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Bleeding-relatedEvent Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of bleeding-related event complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.19 |

## 2.4.20 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant anticoagulant or |
| Statistical Analysis | antiplatelet drugs (Concomitant anticoagulant / antiplatelet , Anticoagulant only, |
| | Antiplatelet only, Neither). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.20 |

# 2.4.21 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence of Concomitant Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile the types of adverse drug reactions (bleeding-related events) by presence or |
| Statistical Analysis | absence of concomitant anticoagulant or antiplatelet drugs (Concomitant |
| | anticoagulant / antiplatelet , Anticoagulant only, Antiplatelet only, Neither). |
| | The compilation method of the types of adverse drug reactions is the same as |
| | described in section 2.4.1. |
| Figure/Table No. | Table 2.4.21 |

#### 2.4.22 Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose fasting |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline fasting triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.22 |

#### 2.4.23 Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose random |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline random triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.23 |

#### 2.4.24 Onset Status of Adverse Drug Reactions or Infections by Initial Dose

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by initial dose. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.24 |

#### 2.4.25 Onset Status of Adverse Drug Reactions or Infections by Breakdown of Change in Daily Dose

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by breakdown of change in daily dose (2 g $\rightarrow$ 4 g, 4 g $\rightarrow$ 2 g, |
| Statistical Analysis | Other). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.25 |

# 2.4.26 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of ConcomitantAntihyperlipidemic Drug Use (during observation period)

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant antihyperlipidemic drug |
| Statistical Analysis | use. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.26 |

# 2.4.27 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of ConcomitantStatins Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant statins drugs. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.27 |

## 2.4.28 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant Fibrate Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant fibrate drugs. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.28 |

## 2.4.29 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant Intestinal Transporter Inhibitors

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant intestinal transporter |
| Statistical Analysis | inhibitors. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.29 |

## 2.4.30 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant Anion-exchange Resin

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant anion-exchange resin. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.30 |

## 2.4.31 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant Nicotinic Acid Derivatives

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant nicotinic acid derivatives. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.31 |

## 2.4.32 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant Probucol

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant probucol. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.32 |

# 2.4.33 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of ConcomitantEthyl Icosapentate (EPA)

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant ethyl icosapentate (EPA). |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.33 |

#### 2.4.34 Changes in Laboratory Test Values (Glucose Metabolism)

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. |
| Figure/Table No. | Table 2.4.34 |

#### 2.4.35 Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. |
| Remarks | Stratification factor: With diabetic complications |
| Figure/Table No. | Table 2.4.35 |

### 2.4.36 Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. |
| Remarks | Stratification factor: Without diabetic complications |
| Figure/Table No. | Table 2.4.36 |

### 2.4.37 Summary of Onset Status of Serious Adverse Events (Exhibit 2-2)

| 2.4.37 Sullillary | of Offset Status of Serious A | diverse Events (Exhibit 2-2) |
|---|---|---|
| Statistical Analysis | Safety-evaluable patients | in clinical studies before approval (total of patients in |
| Set | clinical studies in Japan used for safety evaluation stated in the Adverse Drug | |
| 200 | Reactions section of the pa | ckage insert) and this special drug use surveillance |
| Details of | Compile the following item | ns per survey unit period of the prior-approval status and of |
| Statistical Analysis | the special drug use surveil | llance. |
| Statistical 7 Marysis | Statistical analysis of 'num | nber of study sites,' 'number of surveyed patients,' 'number |
| | - | of SAEs' should cover safety-evaluable patients locked |
| | during each survey unit per | |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients | Number of patients with SAEs |
| | Number of SAEs | Number of SAEs Every PT occurring should be counted as one event. |
| | Rate of patients | Calculated by the following equation: [Number of Patients with SAEs] / [Number of Safety-Evaluable Patients] × 100. |
| | SAE type | The calculation method in performing each analysis should be as follows: [Number of patients with SAEs] • Number of patients in which SAEs occurred. [Number of SAEs] • Number of SAEs that occurred. If the same SAE occurs more than once in the same patient, a total of frequencies of the SAE should be counted. [Rate of patients with SAEs] • Calculated by the following equation: [Number of Patients with SAEs] / [Number of Safety-Evaluable Patients] × 100. [SAE type] • SAEs should be replaced by MedDRA terms. Categorize by SOC and compile SAEs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile SAEs by PT. • At SOC level, the numbers and rates of patients with SAEs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, SAEs should be counted as one patient in the SOC. At PT level, the numbers and rates of patients with SAEs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, SAEs should be counted as one patient in the PT. |

| Figure/Table No. | special drug use surveillance Table 2.4.37 | patients per survey unit period. Do not double-count the same medical institution when counting the number of study sites. |
|---|---|---|
| | Cumulative total of | The number of SAEs of which causal relationship to the Drug has been denied should be entered in the [ ] brackets. In that case, if the same PT events which are both "related" and "not related" in causality to the Drug occur in the same patient, the SAEs should be counted as one patient in the "related" category. A respective total of the numbers of study sites and patients per survey unit period. |

#### 2.4.38 Summary of Onset Status of Serious Adverse Drug Reactions or Infections

| Statistical Analysis | Safety-evaluable patients in | n this special drug use surveillance |
|---|---|---|
| Set | | |
| Details of | Compile the following iten | 1S. |
| Statistical Analysis | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients | Number of patients with serious ADRs |
| | Number of serious<br>ADRs | Number of serious ADRs Every PT occurring should be counted as one event. |
| | Rate of patients | Calculated by the following equation: [Number of Patients with serious ADRs] / [Number of Safety-Evaluable Patients] × 100. |
| | Serious ADR type | The calculation method in performing each analysis should be as follows: [Number of patients with serious ADRs] Number of serious ADRs] Number of serious ADRs that occurred. If the same serious ADR occurs more than once in the same patient, a total of frequencies of the serious ADR should be counted. [Rate of patients with serious ADRs] Calculated by the following equation: [Number of Patients with serious ADRs] / [Number of Safety-Evaluable Patients] × 100. [Serious ADR type] Serious ADRs should be replaced by MedDRA terms. Categorize by SOC and compile serious ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile serious ADRs by PT. At SOC level, the numbers and rates of patients with serious ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, serious ADRs should be counted as one patient in the SOC. At PT level, the numbers and rates of patients with serious ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, serious ADRs should be counted as one patient in the PT. The number of serious ADRs of which causal relationship to the Drug has been denied should be |

| | | entered in the [ ] brackets. In that case, if the same PT events which are both "related" and "not related" in causality to the Drug occur in the same patient, the SAEs should be counted as one patient in the "related" category. |
|---|---|---|
| Figure/Table No. | Table 2.4.38 | |

## 2.4.39 Summary of Onset Status of Serious Adverse Events in Safety-Unevaluable patients

| Statistical Analysis | Safety-unevaluable patients | s in this special drug use surveillance |
|---|---|---|
| Set | | |
| Details of | Compile the following item | |
| Statistical Analysis | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-unevaluable patients. |
| | Number of patients | Number of patients with SAEs |
| | Number of SAEs | Number of SAEs Every PT occurring should be counted as one event. |
| | Rate of patients | Calculated by the following equation: [Number of Patients with SAEs] / [Number of Safety-unevaluable Patients] × 100. |
| | SAE type | The calculation method in performing each analysis should be as follows: [Number of patients with SAEs] • Number of patients in which SAEs occurred. [Number of SAEs] • Number of SAEs that occurred. If the same SAE occurs more than once in the same patient, a total of frequencies of the SAE should be counted. [SAE type] • SAEs should be replaced by MedDRA terms. Categorize by SOC and compile SAEs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile SAEs by PT. • At SOC level, the numbers and rates of patients with SAEs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, SAEs should be counted as one patient in the SOC. At PT level, the numbers of patients with SAEs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, SAEs should be counted as one patient, SAEs should be counted as one patient, SAEs should be counted as one patient, SAEs should be counted as one patient in the PT. |

| | | The number of SAEs of which causal relationship to the Drug has been denied should be entered in the [ ] brackets. In that case, if the same PT events which are both "related" and "not related" in causality to the Drug occur in the same patient, the SAEs should be counted as one patient in the "related" category. |
|---|---|---|
| Figure/Table No. | Table 2.4.39 | |

# 2.4.40 Summary of Onset Status of Serious Adverse Drug Reactions or Infections in Safety-Unevaluable patients

| Statistical Analysis | Safety-unevaluable patients in this special drug use surveillance | | |
|---|---|--|--|
| Set | | | |
| Details of | Compile the following items. | | |
| Statistical Analysis | Item Name Details of Statistical Analysis | | |
| | Number of study sites Number of medical institutions that have collected eCRFs | | |
| | Number of surveyed patients Number of safety-unevaluable patients. | | |
| | Number of patients | | |
| | Number of serious Number of serious ADRs ADRs Every PT occurring should be counted as one event. | | |
| | Rate of patients Calculated by the following equation: [Number of Patients with serious ADRs] / [Number of Safety-unevaluable Patients] × 100. | | |
| | The calculation method in performing each analysis should be as follows: [Number of patients with serious ADRs] • Number of patients in which serious ADRs occurred. [Number of serious ADRs] • Number of serious ADRs that occurred. If the same serious ADR occurs more than once in the same patient, a total of frequencies of the serious ADR should be counted. [Serious ADR type] • Serious ADRs should be replaced by MedDRA terms. Categorize by SOC and compile serious ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile serious ADRs by PT. • At SOC level, the numbers and rates of patients with serious ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, serious ADRs should be counted as one patient in the SOC. At PT level, the numbers of patients with serious | | |
| E' /T.11. N. | T.11. 2.4.40 | ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, serious ADRs should be counted as one patient in the PT. The number of serious ADRs of which causal relationship to the Drug has been denied should be entered in the [ ] brackets. In that case, if the same PT events which are both "related" and "not related" in causality to the Drug occur in the same patient, the serious ADRs should be counted as one patient in the "related" category. |
|---|---|---|
| Figure/Table No. | Table 2.4.40 | |

#### 2.5 Efficacy Statistical Analysis

#### 2.5.1 Changes in Laboratory Test Values (Fasting Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), LDL cholesterol |
| | (Friedewald formula) (mg/dL), VLDL cholesterol (mg/dL), VLDL cholesterol |
| | (%),Apo-B (mg/dL), Apo-CIII (mg/dL), lipoprotein(a) (mg/dL), and remnant |
| | lipoprotein cholesterol (mg/dL). In addition, calculate the 95% confidence interval for |
| | the mean value for rates of change from baseline (%). |
| Figure/Table No. | Table 2.5.1 |

#### 2.5.2 Changes in Laboratory Test Values (Random Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for random measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), VLDL cholesterol |
| | (mg/dL), VLDL cholesterol (%), Apo-B (mg/dL), Apo-CIII (mg/dL), lipoprotein(a) |
| | (mg/dL), and remnant lipoprotein cholesterol (mg/dL). In addition, calculate the 95% |
| | confidence interval for the mean value for rates of change from baseline (%). |
| Figure/Table No. | Table 2.5.2 |

#### 2.5.3 Changes in Laboratory Test Values (Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for random measurements |
| Statistical Analysis | and rates of change from baseline (%) of total cholesterol (mg/dL), LDL cholesterol |
| | (direct measurement) (mg/dL), HDL cholesterol (mg/dL), non-HDL cholesterol |
| | (mg/dL), Apo-AI (mg/dL). In addition, calculate the 95% confidence interval for the |
| | mean value for rates of change from baseline (%). |
| Figure/Table No. | Table 2.5.3 |

# 2.5.4 Changes in Fasting Lipid-Related Ratio

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for TC/HDL-C, |
| Statistical Analysis | LDL-C/HDL-C, and LDL-C/Apo-B. |
| Figure/Table No. Table 2.5.4 | |

# 2.5.5 Changes in Fasting Triglyceride by Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients | in this special drug use surveillance |
|---|---|---|
| Set | | |
| Details of | Calculate summary statisti | ics by stratification for each item for baseline and final |
| Statistical Analysis | evaluation timepoint measu | urements and rates of change from baseline (%) of fasting |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | BMI | Less than 18.5kg/m <sup>2</sup> , 18.5 to less than 25kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Fasting triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |
| | Breakdown of concomitant antihyperlipidemic drugs (during | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |

| | observation period) |
|------------------------------|---------------------|
| Figure/Table No. Table 2.5.5 | ble 2.5.5 |

# 2.5.6 Changes in Random Triglyceride by Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of random | |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | BMI | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |
| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |
| Figure/Table No. | Table 2.5.6 | |

# Statistical Analysis Plan

# (for Periodic Safety Reporting/Reexamination Application)

<Lotriga Granular Capsules>

[Long-term use]

Takeda Pharmaceutical Company Limited Japan Development Center Director of Biostatistics Division



#### Table of Contents

| 1.0 | Defini | tions of Terms | 1 |
|---|---|---|---|
| 1.1 | Def | initions | 1 |
| 1.2 | Nur | nber of Display Digits | 5 |
| 1.3 | Level of Significance | | |
| 1.4 | Handling of Evaluation Timepoint Data | | |
| 2.0 | Result | s of Special Drug Use Surveillance (Survey 1) | 7 |
| 2.1 | Pati | ent Breakdown (Patient Disposition) | 7 |
| 2.2 | Pati | ent Demographics | 8 |
| 2.3 | Trea | atment Details | 10 |
| 2.4 | Safe | ety Statistical Analysis | 12 |
| 2 | .4.1 | Onset Status of Adverse Drug Reactions or Infections (Exhibit 2) | 12 |
| 2 | .4.2 | Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients (Exhibit 2) | 14 |
| 2 | .4.3 | Onset Status of AE | . 15 |
| 2 | .4.4 | Onset Status of Adverse Events in Safety-Unevaluable Patients | . 15 |
| 2 | .4.5 | Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome | :15 |
| 2 | .4.6 | Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome | 16 |
| 2 | .4.7 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Time | me, |
| a | nd Outo | come | 16 |
| 2 | .4.8 | Rate of Patients of Adverse Drug Reactions or Infections by Factor of Patient Demographics | and |
| T | reatme | nt Details | . 17 |
| 2 | .4.9 | Onset Status of Adverse Drug Reactions or Infections by Age Group | 20 |
| 2 | .4.10 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Li | ver |
| C | Complic | ations | 20 |
| 2 | .4.11 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kide | ney |
| C | Complic | ations | 20 |
| 2 | .4.12 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomit | tant |
| A | Anticoag | gulant and/or Antiplatelet Drugs | 20 |
| 2 | .4.13 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence | of |
| C | Concom | itant Anticoagulant and/or Antiplatelet Drugs | 21 |
| 2 | .4.14 | Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level | 21 |
| 2 | .4.15 | Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level | . 21 |
| 2 | .4.16 | Changes in Laboratory Test Values (Glucose Metabolism) | . 21 |
| 2 | .4.17 | Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications> | . 22 |
| 2 | .4.18 | Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications> | 22 |
| 2.5 | Effi | cacy Statistical Analysis | 23 |
| 2 | .5.1 | Changes in Laboratory Test Values (Fasting Lipid) | 23 |
| 2 | .5.2 | Changes in Laboratory Test Values (Random Lipid) | 23 |

| | 2.5.3 | Changes in Fasting Lipid-Related Ratio. | 23 |
|---|---|---|---|
| | 2.5.4 | Changes in Fasting Triglyceride by Factor of Patient Demographics and Treatment Details | 24 |
| | 2.5.5 | Changes in Random Triglyceride by Factor of Patient Demographics and Treatment Details | 25 |
| 3.0 | Summa | ary of Onset Status of Serious Adverse Events (Exhibit 2-2) | 26 |

#### 1.0 Definitions of Terms

# 1.1 Definitions

| Item | Definition |
|---|---|
| Survey unit period | Periodic Safety Report 1: July 22, 2012 to January 21, 2013 |
| (periodic safety report) | Periodic Safety Report 2: January 22, 2013 to July 21, 2013 |
| | Periodic Safety Report 3: July 22, 2013 to January 21, 2014 |
| | Periodic Safety Report 4: January 22, 2014 to July 21, 2014 |
| | Periodic Safety Report 5: July 22, 2014 to July 21, 2015 |
| | Periodic Safety Report 6: July 22, 2015 to July 21, 2016 |
| | Periodic Safety Report 7: July 22, 2016 to July 21, 2017 |
| Drug | Lotriga Granular Capsules |
| SOC | System organ class of MedDRA. |
| HLGT | High level group term of MedDRA. |
| PT | Preferred term of MedDRA. |
| LLT | Lowest level term of MedDRA. |
| Enrolled patient | A patient approved for enrollment in the Study. |
| Patient with eCRF | An enrolled patient whose eCRF was submitted via |
| collected | |
| Patient with eCRF | An enrolled patient other than a patient with eCRF collected. |
| uncollected | |
| Locked patient | A patient who has completed the approval process in the PMS system. |
| Unlocked patient | A patient with eCRF collected other than a locked patient. |
| Safety-evaluable patient | A locked patient included in safety evaluation. |
| Safety-unevaluable patient | A locked patient excluded from safety evaluation. |
| Efficacy-evaluable patient | A safety-evaluable patient included in efficacy evaluation. |
| Efficacy-unevaluable | A safety-evaluable patient excluded from efficacy evaluation. |
| patient | |
| ADR | An abbreviated form of the term 'adverse drug reaction or infection.' |
| | Refers to an adverse event other than those judged by the investigator as 'not |
| | related' in causality to the Drug. |
| | In this plan, 'adverse drug reactions or infections' is used in headings, and |
| | 'ADRs' is used in the text and tables. |
| Serious adverse event | [Prior-approval data] |
| (SAE) | An adverse event (AE) judged as 'serious' by the trial investigator. |
| | [Surveillance data] |
| | An adverse event (AE) judged as 'serious' by the investigator. |
| | Note that events listed in the separate MedDRA code list of the Takeda |
| | Medically Significant AE List should be treated as serious even if judged as |
| | 'not serious' by the investigator. |

| Item | Definition |
|---|---|
| Bleeding-related event | An event falling under Standardized MedDRA Query (SMQ) code 20000038 |
| | (hemorrhagic SMQ [narrow scope]). |
| Rate of patients | [For safety compilation with safety-evaluable patients] |
| | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Evaluable Patients] × 100. |
| | [For safety compilation with safety-unevaluable patients] |
| | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Unevaluable Patients] × 100. |
| Incidence | [For safety compilation with safety-evaluable patients] |
| | Calculated by the following equation: [Number of Events] / [Number of |
| | Safety-Evaluable Patients] × 100. |
| | [For safety compilation with safety-unevaluable patients] |
| | Calculated by the following equation: [Number of Events] / [Number of |
| | Safety-Unevaluable Patients] × 100. |
| Onset time | Calculated by the following equation: [Onset Date] - [Start Date] + 1. |
| | If the onset date is unknown, use the first day of the month as the onset date in |
| | this equation. However, use the start date as the onset date if [Start Year & |
| | Month] = [Onset Year & Month]. |
| Liver patient | A patient with 'fatty liver,' 'alcoholic fatty liver,' 'chronic hepatitis' or 'hepatic |
| | cirrhosis' check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SMQ code 20000005 (hepatic SMQ [narrow |
| | scope]) in the Complication Details (Other Diseases) field. |
| Kidney patient | A patient with 'diabetic nephropathy,' 'glomerulonephritis' or 'chronic kidney |
| | disease (CKD)' check-marked in the Complication Details field. Or a patient |
| | with a complication falling under the Takeda MedDRA query (TMQ) (Renal |
| | Disease) in the Complication Details (Other Diseases) field. |
| Heart patient | A patient with 'myocardial infarction,' 'angina pectoris' or 'atrial fibrillation' |
| | check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SOC code 10007541 (cardiac disorders) in the |
| | Complication Details (Other Diseases) field. |
| Cerebrovascular patient | A patient with 'cerebral infarction' or 'cerebral hemorrhage' check-marked in |
| | the Complication Details field. Or a patient with a complication falling under |
| | the SMQ code 20000060 (cerebrovascular SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Diabetic patient | A patient with 'diabetes' check-marked in the Complication Details field. Or a |
| | patient with a complication falling under the TMQ code (Diabetes Mellitus |
| | Confirmed diagnosis, excl diagnostics) in the Complication Details (Other |
| | Diseases) field. |

| Item | Definition |
|---|---|
| Hypertensive patient | A patient with 'hypertension' check-marked in the Complication Details field. |
| | Or a patient with a complication falling under the SMQ code 20000147 |
| | (hypertensive SMQ [narrow scope]) in the Complication Details (Other |
| | Diseases) field. |
| Myocardial infarction | A patient with 'myocardial infarction' check-marked in the Complication |
| patient | Details field. Or a patient with a complication falling under the SMQ code |
| | 20000047 (myocardial infarction SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Anginal patient | A patient with 'angina pectoris' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10002383 (angina pectoris), 10002388 (unstable angina pectoris), 10036759 |
| | (Prinzmetal angina), or 10058144 (postinfarction angina) in the Complication |
| | Details (Other Diseases) field. |
| Atrial fibrillation patient | A patient with 'atrial fibrillation' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10003658 (atrial fibrillation) in the Complication Details (Other Diseases) |
| | field. |
| Ischemic cerebrovascular | A patient with 'cerebral infarction' check-marked in the Complication Details |
| patient | field. Or a patient with a complication falling under the SMQ code 2000000 |
| | (ischemic cerebrovascular disease SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Hemorrhagic | A patient with 'cerebral hemorrhage' check-marked in the Complication Detail |
| cerebrovascular patient | field. Or a patient with a complication falling under the SMQ code 20000064 |
| | (hemorrhagic cerebrovascular disease SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Bleeding-related event | A patient with a complication falling under the SMQ code 20000038 (bleeding |
| patient | SMQ [narrow scope]) in the Complication Details (Other Diseases) field. |
| Age | Calculated by the following equation: [Start Year] - [Birth Year] - 1 if [Start |
| | Month & Day] < [Birth Month & Day]. |
| | Calculated by the following equation: [Start Year] - [Birth Year] if [Start Month |
| | & Day] ≥ [Birth Month & Day]. |
| | If the birth day is unknown, use the first day of the month instead in this |
| DMI | equation. Calculated by the following equation: [Weight (leg)] / (0,0001 × [Height (am)]) |
| BMI | Calculated by the following equation: [Weight (kg)] / (0.0001 × [Height (cm)] |
| Diament and | × [Height (cm)]). Indicated by rounding off to the first decimal place. |
| Disease duration (in years) | Calculated by the following equation: ([Start Year & Month] - [Year & Month] |
| | of Hyperlipidemia Diagnosis] + 1) / 12. Indicated by rounding off to the first |
| | decimal place. |

| Item | Definition |
|---|---|
| Start date | The start date of first administration of the Drug stated in the Treatment |
| | Duration field of the eCRF. |
| End date | The end date of last administration of the Drug stated in the Treatment Duration |
| | field of the eCRF. |
| | However, if the end date of last administration is in 'ongoing 12 months after |
| | baseline,' the end date should be the start date plus 405 days. |
| Observation period (in | Refers to the entire period of observation. The start date and end date of |
| days) | observation period should be the same as the 'start date' and 'end date,' |
| | respectively. Calculated by the following equation: [End Date] - [Start |
| | Date] + 1. |
| Treatment duration (in | Refers to the entire period of treatment. A total of Drug dosing periods in the |
| days) | number of actual administration days, excluding washout period. Calculated as |
| | a total of ([End Date] - [Start Date] + 1) in the number of actual administration |
| | days, excluding washout period. |
| Mean daily dose | Calculated by the following equation: Total of ([Daily Dose] × [Total Period of |
| | Treatment with the Dose]) / [Observation Period]. See the above for calculation |
| | of observation period. |
| Concomitant medication | A drug used during the surveillance period. However, concomitant medications |
| | exclude drugs used for adverse events occurring during the period. |
| Antihyperlipidemic drug | A drug starting with any of the following drug codes: 218, 2190006, 2190101, |
| | 2190102, 2190103, 2190104, 290006, 3133001, 3133400, 3399004. |
| Statins drug | A drug starting with any of the following drug codes: 2189010, 2189011, |
| | 2189012, 2189015, 2189016, 2189017. |
| Fibrate drug | A drug starting with drug code: 2183. |
| Intestinal transporter | A drug starting with drug code: 2189018. |
| inhibitor | |
| Anion-exchange resin | A drug starting with any of the following drug codes: 2189009, 2189014. |
| Nicotinic acid derivative | A drug starting with any of the following drug codes: 2189004, 2189005, |
| | 2190006. |
| Probucol | A drug starting with drug code: 2189008. |
| Ethyl icosapentate (EPA) | A drug starting with drug code: 3399004. |
| Anticoagulant drug | A drug starting with any of the following drug codes: 333, 2190408, 6343424. |
| Antiplatelet drug | A drug starting with any of the following drug codes: 3399 (excluding |
| | 3399004), 2171010, 2171402. |
| Anticoagulant/antiplatelet | A drug that falls under the class of either anticoagulant or antiplatelet drugs |
| drug | |

| Item | Definition |
|---|---|
| LDL cholesterol | Calculated the equation below if the patient is fasting at the time of blood |
| (Friedewald formula) | collection for laboratory testing with triglyceride 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol - triglyceride / 5 |
| Non-HDL cholesterol | Calculated by the equation below if triglyceride is 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol |
| TC/LDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | Total cholesterol / LDL cholesterol (Friedewald formula) |
| LDL-C/HDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / HDL cholesterol |
| LDL-C/Apo-B ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / Apo-B |
| Summary statistics | Mean value, standard deviation, minimum value, first quartile, median, third |
| | quartile, maximum value |

# 1.2 Number of Display Digits

| Item | Definition |
|---|---|
| Percentage (%) | Rate of patients with ADRs: |
| | Indicated by rounding off to the second decimal place. |
| | Other than above: |
| | Indicated by rounding off to the first decimal place. |
| Summary statistics | Mean value: |
| | Indicated by rounding off to the first digit below the raw numerical data. |
| | Standard deviation: |
| | Indicated by rounding off to the second digit below the raw numerical data. |
| | First quartile, median, third quartile: |
| | Indicated by rounding off to the first digit below the raw numerical data. |
| | Minimum value, maximum value: |
| | Indicated at the same digits of the raw numerical data. |
| Confidence interval | Indicated by rounding off to the second digit below the raw numerical data. |

# 1.3 Confidence Coefficient

Two-sided 95%

#### 1.4 Handling of Evaluation Timepoint Data

The evaluation timepoints are the start of treatment with the Drug (baseline), Month 3, Month 6, Month 9, Month 12, and final evaluation timepoint.

If multiple data exist within each evaluation timepoint, calculate absolute values of difference in measurement intervals from the basic day count and adopt the minimum absolute value as date for that evaluation timepoint. If all the absolute values are the same, adopt one for the latest date of testing/measurement. Test/Measurement values should not be adopted that have been obtained after completion of treatment with the Drug. The final evaluation timepoint test/measurement should be one taken on the latest date within 405 days elapsed since the start date (including values tested/measured during washout period). Note that the number days elapsed since the start date should be counted with the start date as day 0 and the previous day as day -1.

| Evaluation Timepoint | Tolerance (Number of Days Since Baseline) | Basic Day Count |
|---|---|---|
| Baseline | -90 to 0 | 0 |
| Month 3 | 1 to 135 | 90 |
| Month 6 | 136 to 225 | 180 |
| Month 9 | 226 to 315 | 270 |
| Month 12 | 316 to 405 | 360 |
| Final evaluation | 1 to 405 | - |
| timepoint | | |

#### 2.0 Results of Special Drug Use Surveillance (Survey 1)

<Lotriga Granular Capsules Special Drug Use Surveillance [long-term use survey]>

# 2.1 Patient Breakdown (Patient Disposition)

| Statistical Analysis | Enrolled patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Number of enrolled patients, number of patient enrollment sites, number of patients |
| Statistical Analysis | with eCRFs collected, number of patients with eCRFs uncollected, number of loc |
| | patients, number of unlocked patients, number of safety-evaluable patients, number of |
| | safety-unevaluable patients, number of efficacy-evaluable patients, number of |
| | efficacy-unevaluable patients |
| | Do not double-count the same medical institution with different participating clinical |
| | departments when counting the number of patient enrollment sites. |
| | Count the number of patients per reason below for not collecting and total the |
| | numbers when the number of patients with eCRFs uncollected. |
| | <reasons collecting="" for="" not=""></reasons> |
| | Survey under way |
| | • eCRFs uncollectable |
| | Investigator transferred |
| | Investigator's health reasons |
| | Patients enrolled 15 days after Drug prescription [before eCRF collection] |
| | • Others |
| | Count the number of patients per reason below for exclusion and total the numbers |
| | when counting the numbers of safety- and efficacy-unevaluable patients. If the same |
| | patient falls under multiple reasons for exclusion, they should be counted separately. |
| | <reasons evaluation="" exclusion="" for="" from="" safety=""></reasons> |
| | Drug administered before contract period |
| | Patient enrolled 15 days after Drug prescription |
| | No data available after Drug administration |
| | Drug not administered |
| | <reasons efficacy="" evaluation="" exclusion="" for="" from=""></reasons> |
| | Pre- or post-administration lipid-related values (fasting or random) unavailable |
| | No output needs to be generated for items for which the number of patients is zero. |
| | For periodic safety reports, the numbers of efficacy-evaluable and unevaluable |
| | patients should not be counted. |
| Figure/Table No. | Figure 2.1, Table 2.1 |

# 2.2 Patient Demographics

| Statistical Analysis<br>Set | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Details of<br>Statistical Analysis | Categorize the patient population by the following categories for each item and compile the number of patients and incidence. | |
| Š | Item Name | Category |
| | Sex | Male, Female |
| | Age | Summary statistics |
| | | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | Treatment category | Outpatient, inpatient |
| | BMI | Summary statistics |
| | | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | | Hypertension, Diabetic, Liver disorder, Kidney |
| | | disorder, Cardiac disorders [myocardial infarction, |
| | Complication | angina pectoris, atrial fibrillation, others], |
| | breakdown | Cerebrovascular diseases [hemorrhagic |
| | | cerebrovascular disease, ischemic cerebrovascular |
| | | disease, others], Bleeding-related event, Others |
| | Drinking history | |
| | (Does the patient | |
| | drink alcoholic | Yes, No, Unknown |
| | beverages nearly | |
| | every day?) | |
| | | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | | to less than 500 mg/dL, 500mg/dL or over, Not |
| | Fasting triglyceride a | t measured |
| | baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 |
| | | to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | | 750 mg/dL or over, Not measured |
| | | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | | to less than 500 mg/dL, 500mg/dL or over, Not |
| | Random triglyceride | measured |
| | at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 |
| | | to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | | 750 mg/dL or over, Not measured |

| | Smoking history | Never, Current, Former, Unknown |
|---|---|---|
| | Hypersensitivity disposition | No, Yes, Unknown |
| | | Summary statistics |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence of surgery within one month before baseline | No, Yes |
| | Pregnancy status during treatment (only for female) | No, Yes |
| Figure/Table No. | Table 2.2 | |

#### 2.3 Treatment Details

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of<br>Statistical Analysis | Categorize the patient population by the following categories for each item and compile the number of patients and incidence. | |
| | Item Name | Category |
| | Initial dose | 2 g, 4 g, Other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |
| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | Statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others |
| | Presence or absence of concomitant anticoagulant/antiplatelet drug use (during observation period) | No, Yes |
| | Breakdown of concomitant anticoagulant/antiplatelet drugs (during observation period) | Anticoagulant drugs, antiplatelet drugs |
| | Completion of treatment with the Drug | No, Yes, Unknown |

| | Reason for treatment | Treatment goal achieved, AE developing, Patient no |
|---|---|---|
| | completion | longer visiting hospital due to hospital transfer or |
| | | otherwise, Insufficient effect, Other |
| Figure/Table No. | Table 2.3 | |

# 2.4 Safety Statistical Analysis

# 2.4.1 Onset Status of Adverse Drug Reactions or Infections (Exhibit 2)

| Ctatistical Assalassia | Cafata analas la matianta in | -lining -t-lin - 1-f |
|---|---|---|
| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in | |
| Set | clinical studies in Japan used for safety evaluation stated in the Adverse Drug | |
| | Reactions section of the package insert) and this special drug use surveillance | |
| Details of | Compile the following items for the prior-approval status and per survey unit period | |
| Statistical Analysis | of the special drug use survei | llance. |
| | Statistical analysis of 'number | er of study sites,' 'number of surveyed patients,' 'number |
| | of patients with ADRs,' and | 'number of ADRs' should cover safety-evaluable patients |
| | locked during each survey ur | nit period. |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients with ADRs | Number of patients in which ADRs occurred. |
| | | Number of ADRs that occurred. |
| | Number of ADRs | Every PT occurring should be counted as one event. |
| | D ( C ( ) ( ) | Calculated by the following equation: [Number of |
| | Rate of patients with ADRs | Patients with ADRs] / [Number of |
| | | Safety-Evaluable Patients] × 100 |
| | | The calculation method in performing each analysis should be as follows: |
| | | [Number of patients with ADRs] |
| | | Number of patients in which ADRs occurred. |
| | | [Number of ADRs] • Number of ADRs that occurred. If the same ADR |
| | | occurs more than once in the same patient, a total of frequencies of the ADR should be counted. |
| | | [Rate of patients with ADRs] |
| | | • Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Evaluable Patients] × 100. |
| | ADD 4 | [ADR type] |
| | ADR type | • ADRs should be replaced by MedDRA terms. |
| | | Categorize by SOC and compile ADRs by PT in |
| | | each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order |
| | | but without outputting) and compile ADRs by PT. |
| | | • At SOC level, the numbers and rates of patients |
| | | with ADRs should be presented by SOC |
| | | internationally agreed order. If the same SOC |
| | | occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. |
| | | At PT level, the numbers and rates of patients with |
| | | ADRs should be presented by PT code in |

| | Cumulative total for special drug use surveillance | ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the PT. A respective total of the numbers of study sites and patients per survey unit period. Do not double-count the same medical institution when counting the number of study sites. |
|---|---|---|
| Figure/Table No. | Table 2.4.1 | |

# 2.4.2 Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients

| Set clinical studies inside and outside Japan used for safety evaluation stated in the Adverse Drug Reactions section of the package insert) and this specified drug use surveillance Details of Statistical Analysis Time Name | Statistical Analysis | Safety-unevaluable natients i | in clinical studies before approval (total of natients in |
|---|---|---|---|
| Adverse Drug Reactions section of the package insert) and this specified drug use surveillance Details | | Safety-unevaluable patients in clinical studies before approval (total of patients in | |
| Details of Statistical Analysis Item Name | Set | - | |
| Compile the following items. | | | |
| Statistical Analysis Number of study sites Number of medical institutions that have collected cCRFs Number of surveyed patients Number of safety-unevaluable patients Number of patients with ADRs Number of ADRs that have occurred. Number of ADRs Number of ADRs that have occurred. Number of ADRs Every PT occurring should be counted as one event. Rate of patients with ADRs Number of Patients with ADRs Number of Safety-Unevaluable Patients] × 100 The calculation method in performing each analysis should be as follows: [Number of Patients with ADRs] Number of Patients in which ADRs occurred. [Number of Patients in which ADRs occurred. [Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] Number of Safety-Unevaluable Patients] × 100. ADR type ADRs should be replaced by MedDRA terms. ADR type ADRs should be replaced by MedDRA terms. ADR should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers and rates of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted | D + 11 C | | |
| Number of surveyed patients Number of surveyed patients Number of patients with ADRs Number of ADRs Number of ADRs that have occurred. Number of Safety-Unevaluable Patients] × 100 The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] • Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] • ADRs should be replaced by MedDRA terms. Categories by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC. At PT level, the numbers and rates of patients with ADRs should be counted as one patient in the SOC. | | | Date la constitución de la constitución |
| Number of surveyed patients Number of patients with ADRs Number of ADRs Number of ADRs burney PT occurring should be counted as one event. Rate of patients with ADRs Calculated by the following equation: [Number of Patients with ADRs] Number of ADRs Calculated by the following equation: [Number of Patients with ADRs] Number of patients with ADRs] Number of patients with ADRs] Number of patients with ADRs] Number of Patients with ADRs] Number of Patients with ADRs occurred. [Number of Patients with ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] Calculated by the following equation: [Number of ADRs that occurred.] Number of Patients with ADRs occurred. [Number of ADRs that occurred.] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] Calculated by the following equation: [Number of Patients with ADRs] ADR type ADR type [1] ADR should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. | Statistical Analysis | | |
| Number of patients with ADRs Number of ADRs Number of ADRs that have occurred. Number of ADRs that have occurred. Every PT occurring should be counted as one event. Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100 The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] • Number of patients in which ADRs occurred. [Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] • Calculated by the following equation: [Number of Safety-Unevaluable Patients] × 100. [ADR type] • ADR should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers and rates of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. | | Number of study sites | |
| Number of ADRs Number of ADRs that have occurred. Every PT occurring should be counted as one event. Rate of patients with ADRs / [Number of Patients with ADRs] / [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100 The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] Number of patients in which ADRs occurred. [Number of ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] Calculated by the following equation: [Number of Patients with ADRs] Calculated by the following equation: [Number of Patients with ADRs] / [Number of Patients with ADRs] / [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100. [ADR type] ADR should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers and rates of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. | | patients | Number of safety-unevaluable patients. |
| Rate of patients with ADRs Rate of patients with ADRs Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100 The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] • Number of patients in which ADRs occurred. [Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] • Calculated by the following equation: [Number of Safety-Unevaluable Patients] × 100. [ADR type] • ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient with ADRs should be counted as one patient in the SOC. | | _ | Number of patients in which ADRs occurred. |
| Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100 The calculation method in performing each analysis should be as follows: [Number of patients with ADRs] • Number of patients in which ADRs occurred. [Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100. [ADR type] • ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same PT occurs more than once in the same PT occurs more than once in the same PT occurs more than once in the same patient, ADRs should be counted | | Number of ADRs | Every PT occurring should be counted as one |
| analysis should be as follows: [Number of patients with ADRs] • Number of patients in which ADRs occurred. [Number of ADRs] • Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] • Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100. [ADR type] • ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. • At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be counted as one patient in the SOC. At PT level, the numbers and rates of patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same PT occurs more than once in the same patient, ADRs should be counted as one patient with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted as one patient with ADRs should be counted as one patient with ADRs should be counted by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted by PT code in ascending order. | | _ | Patients with ADRs] / [Number of |
| Figure/Table No. Table 2.4.2 | Figure/Table No. | | analysis should be as follows: [Number of patients with ADRs] Number of patients in which ADRs occurred. [Number of ADRs] Number of ADRs that occurred. If the same ADR occurs more than once in the same patient, a total of frequencies of the ADR should be counted. [Rate of patients with ADRs] Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100. [ADR type] ADRs should be replaced by MedDRA terms. Categorize by SOC and compile ADRs by PT in each category. If SOC is 'Investigations,' classify by HLGT (sort by HLGT code in ascending order but without outputting) and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. If the same SOC occurs more than once in the same patient, ADRs should be presented by PT code in ascending order. If the same SOC occurs more than once in the same patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patients with ADRs should be presented by PT code in ascending order. If the same PT occurs more than once in the same patient, ADRs should be counted |
| Figure/Table No. Table 2.4.2 | Figure/Table No. | Table 2.4.2 | , |

#### 2.4.3 Onset Status of AE

| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in |
|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the |
| | Adverse Drug Reactions section of the package insert) and this special drug use |
| | surveillance |
| Details of | The compilation method is the same as described in section 2.4.1. However, adverse |
| Statistical Analysis | drug reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.3 |

#### 2.4.4 Onset Status of Adverse Events in Safety-Unevaluable Patients

| Statistical Analysis | Safety-unevaluable patients in clinical studies before approval (total of patients in |
|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the |
| | Adverse Drug Reactions section of the package insert) and this specified drug use |
| | surveillance |
| Details of | Compilation method is the same as described in section 2.4.2. However, adverse drug |
| Statistical Analysis | reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.4 |

#### 2.4.5 Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADI | Rs by the following categories for each item and compile ADR types. |
| Statistical Analysis | Item Name | Details of Statistical Analysis |
| | Number of patients | Compile the number of patients with ADRs. |
| | Number of ADRs | At SOC, the number of ADRs should be compiled by totaling associated PTs that occurred. At PT level, every PT occurring should be counted as one event. |
| | Item Name | Category |
| | Seriousness | Serious, Not serious |
| | Onset time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over, Unknown |
| | Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, Death, Unknown |
| Figure/Table No. | Table 2.4.5 | |

#### 2.4.6 Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize AEs | by the following categories for each item and compile AE types. |
| Statistical Analysis | The compilation | on method of AE types is the same as described in section 2.4.5. |
| | However, adver | rse drug reactions should be replaced by adverse events. |
| | Item Name | Category |
| | Seriousness | Serious, Not serious |
| | On got time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to |
| | Onset time | 360 days, 361 days or over, Unknown |
| | Outcomo | Resolved, Resolving, Not resolved, Resolved with sequelae, |
| | Outcome | Death, Unknown |
| | Causal | Causal Related, Not related, Unevaluable |
| | relationship | If AEs (LLTs) occur more than once in the same patient, they |
| | with the | should be counted as one event in the following order of priority: |
| | Drug | (1) Related, (2) Unevaluable, (3) Not related |
| Figure/Table No. | Table 2.4.6 | |

#### 2.4.7 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Time,

#### and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Categorize adverse drug reactions (bleeding-related events) by the following |
| Statistical Analysis | categories for each item, and count the types of adverse drug reactions |
| | (bleeding-related events). |
| | The categories and the compilation method of adverse drug reactions are the same as |
| | described in section 2.4.5. |
| Figure/Table No. | Table 2.4.7 |

# 2.4.8 Rate of Patients of Adverse Drug Reactions or Infections by Patient Demographics and TreatmentDetails

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADRs by the following categories for each item and compile the rate of | |
| Statistical Analysis | patients with ADRs (point estimate and 95% confidence interval). | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | BMI | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | Complication breakdown | Hypertension, Diabetic, Liver disorder, Kidney disorder, Cardiac disorders [myocardial infarction, angina pectoris, atrial fibrillation, others], Cerebrovascular diseases [hemorrhagic cerebrovascular disease, ischaemic cerebrovascular disease, others], Bleeding-related event, Others |
| | Drinking history (Does<br>the patient drink<br>alcoholic beverages<br>nearly every day?) | Yes, No, Unknown |
| | Fasting triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Smoking history | Never, Current, Former, Unknown |

| | Hypersensitivity disposition | No, Yes, Unknown |
|---|---|---|
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence of surgery within one month before baseline | No, Yes |
| | Pregnancy status during treatment (only for female) | No, Yes |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |
| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | Statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others |
| | Presence or absence of concomitant anticoagulant/antiplatelet drug use (during observation period) | No, Yes |
| | Breakdown of concomitant anticoagulant/antiplatelet drugs (during observation period) | Anticoagulant drugs, antiplatelet drugs |
| Figure/Table No. | Table 2.4.8 | |

#### 2.4.9 Onset Status of Adverse Drug Reactions or Infections by Age Group

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Classify the patient population into 64 years or below, 65 to 74 years, and 75 years or |
| Statistical Analysis | over, and compile ADR types. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.9 |

### 2.4.10 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Liver

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of liver complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.10 |

#### 2.4.11 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kidney

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of kidney complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.11 |

# 2.4.12 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant

#### Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant anticoagulant and/or |
| Statistical Analysis | antiplatelet drugs (Both, Anticoagulant only, Antiplatelet only, Neither). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.12 |

# 2.4.13 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence of Concomitant Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile the types of adverse drug reactions (bleeding-related events) by presence or |
| Statistical Analysis | absence of concomitant anticoagulant and/or antiplatelet drugs (Both, Anticoagulant |
| | only, Antiplatelet only, Neither). |
| | The compilation method of the types of adverse drug reactions is the same as |
| | described in section 2.4.1. |
| Figure/Table No. | Table 2.4.13 |

#### 2.4.14 Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose fasting |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline fasting triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.14 |

#### 2.4.15 Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose random |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline random triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.15 |

#### 2.4.16 Changes in Laboratory Test Values (Glucose Metabolism)

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. |
| Figure/Table No. | Table 2.4.16 |

#### 2.4.17 Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. |
| Remarks | Stratification factor: With diabetic complications |
| Figure/Table No. | Table 2.4.17 |

#### 2.4.18 Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. |
| Remarks | Stratification factor: Without diabetic complications |
| Figure/Table No. | Table 2.4.18 |

# 2.5 Efficacy Statistical Analysis

#### 2.5.1 Changes in Laboratory Test Values (Fasting Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), total cholesterol |
| | (mg/dL), LDL cholesterol (direct measurement) (mg/dL), LDL cholesterol |
| | (Friedewald formula) (mg/dL), HDL cholesterol (mg/dL), non-HDL cholesterol |
| | (mg/dL), VLDL cholesterol (mg/dL), VLDL cholesterol (%), Apo-AI (mg/dL), Apo-B |
| | (mg/dL), Apo-CIII (mg/dL), lipoprotein(a) (mg/dL), and remnant lipoprotein |
| | cholesterol (mg/dL). In addition, calculate the 95% confidence interval for the mean |
| | value for rates of change from baseline (%). |
| Figure/Table No. | Table 2.5.1 |

# 2.5.2 Changes in Laboratory Test Values (Random Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom random |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for random measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), total cholesterol |
| | (mg/dL), LDL cholesterol (direct measurement) (mg/dL), HDL cholesterol (mg/dL), |
| | non-HDL cholesterol (mg/dL), VLDL cholesterol (mg/dL), VLDL cholesterol (%) |
| | Apo-AI (mg/dL), Apo-B (mg/dL), Apo-CIII (mg/dL), lipoprotein(a) (mg/dL), and |
| | remnant lipoprotein cholesterol (mg/dL). In addition, calculate the 95% confidence |
| | interval for the mean value for rates of change from baseline (%). |
| Figure/Table No. | Table 2.5.2 |

#### 2.5.3 Changes in Fasting Lipid-Related Ratio

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for TC/LDL-C, |
| Statistical Analysis | LDL-C/HDL-C, and LDL-C/Apo-B. |
| Figure/Table No. | Table 2.5.3 |

#### 2.5.4 Changes in Fasting Triglyceride by Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting | |
|---|---|---|
| Set | blood collection was performed at baseline | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of fasting | |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | BMI | Less than 18.5kg/m <sup>2</sup> , 18.5 to less than 25kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Fasting triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use | |
| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives. Probucol Ethyl icosapentate (EPA) |
| Figure/Table No. | Table 2.5.4 | |

# 2.5.5 Changes in Random Triglyceride by Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom random | |
|---|---|---|
| Set | blood collection was performed at baseline | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of random | |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | ВМІ | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Presence or absence of concomitant antihyperlipidemic drug use (during observation period) | No, Yes |
| | Breakdown of concomitant antihyperlipidemic drugs (during observation period) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |
| Figure/Table No. | Table 2.5.5 | |

#### 3.0 Summary of Onset Status of Serious Adverse Events (Exhibit 2-2)

| | <b>I</b> | , |
|---|---|---|
| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in | |
| Set | clinical studies in Japan used for safety evaluation stated in the Adverse Drug | |
| | Reactions section of the package insert) and this special drug use surveillance | |
| Details of | Compile the following items per survey unit period of the prior-approval status and of | |
| Statistical Analysis | the special drug use surve | illance. |
| Statistical Final yold | Statistical analysis of 'nur | mber of study sites,' 'number of surveyed patients,' 'number |
| | - | r of SAEs' should cover safety-evaluable patients locked |
| | during each survey unit period. | |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients | Number of patients with SAEs |
| | Number of SAEs | Number of SAEs |
| | Number of SAES | Every PT occurring should be counted as one event. |
| | | Calculated by the following equation: [Number of |
| | Rate of patients | Patients with SAEs] / [Number of Safety-Evaluable |
| | Rate of patients | Patients] × 100. |
| | | The calculation method in performing each analysis |
| | | should be as follows: |
| | | [Number of patients with SAEs] |
| | | • Number of patients in which SAEs occurred. |
| | | [Number of SAEs] |
| | | • Number of SAEs that occurred. If the same SAE |
| | | occurs more than once in the same patient, a total of frequencies of the SAEs should be counted. |
| | | [Rate of patients with SAEs] |
| | | • Calculated by the following equation: [Number of Patients with SAEs] / [Number of Safety-Evaluable Patients] × 100. |
| | | [SAE type] |
| | | • SAEs should be replaced by MedDRA terms. |
| | SAE type | Categorize by SOC and compile SAEs by PT in each |
| | Si iii type | category. If SOC is 'Investigations,' classify by HLGT |
| | | (sort by HLGT code in ascending order but without |
| | | outputting) and compile SAEs by PT. |
| | | • At SOC level, the numbers and rates of patients with |
| | | SAEs should be presented by SOC internationally |
| | | agreed order. If the same SOC occurs more than once in the same patient, SAEs should be counted as one patient in the SOC |
| | | patient in the SOC. |
| | | At PT level, the numbers and rates of patients with SAEs should be presented by PT code in ascending |
| | | order. If the same PT occurs more than once in the |
| | | same patient, SAEs should be counted as one patient |
| | | in the PT. |
| | <u> </u> | III UIC 1 1. |

| Figure/Table No. | special drug use surveillance Table 3.0 | Do not double-count the same medical institution when counting the number of study sites. |
|---|---|---|
| | Cumulative total of | patients per survey unit period. |

# Statistical Analysis Plan

# (for Periodic Safety Reporting/Reexamination Application)

# <Lotriga Granular Capsules>

[Long-term use]

Takeda Pharmaceutical Company Limited
Pharmacovigilance Department, Japan Development Center
Postmarketing Surveillance Group Manager

| PPD |
|-----|

Statistical Analysis Contractor



#### Table of Contents

| 1.0 | Defini | tions of Terms | . 1 |
|---|---|---|---|
| 1.1 | Defi | initions | . 1 |
| 1.2 | Nun | nber of Display Digits | . 5 |
| 1.3 | Leve | el of Significance | . 5 |
| 1.4 | Han | dling of Evaluation Timepoint Data | . 6 |
| 2.0 | Result | s of Special Drug Use Surveillance (Survey 1) | . 7 |
| 2.1 | Pati | ent Breakdown (Patient Disposition) | . 7 |
| 2.2 | Pati | ent Demographics | . 8 |
| 2.3 | Trea | ntment Details | 10 |
| 2.4 | Safe | ety Statistical Analysis | 11 |
| 2. | .4.1 | Onset Status of Adverse Drug Reactions or Infections (Exhibit 2) | 11 |
| 2. | .4.2 | Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients (Exhibit 2) | 12 |
| 2. | .4.3 | Onset Status of AE | 12 |
| 2.4.4 Onset Status of Adverse E | | Onset Status of Adverse Events in Safety-Unevaluable Patients | 13 |
| 2. | .4.5 | Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome | 13 |
| 2. | .4.6 | Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome | 14 |
| 2. | .4.7 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Tin | ne, |
| aı | nd Outc | ome | 14 |
| 2. | .4.8 | Rate of Patients of Adverse Drug Reactions or Infections by Factor of Patient Demographics a | nd |
| T | reatmer | nt Details | 15 |
| 2. | .4.9 | Onset Status of Adverse Drug Reactions or Infections by Age Group | 17 |
| 2. | .4.10 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Liv | /er |
| C | omplica | ations | 17 |
| 2. | .4.11 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kidn | ey |
| C | omplica | ations | 17 |
| 2. | .4.12 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomita | ınt |
| A | nticoag | ulant and/or Antiplatelet Drugs | 17 |
| 2. | .4.13 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence | of |
| C | oncomi | tant Anticoagulant and/or Antiplatelet Drugs | 18 |
| 2. | .4.14 | Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level | 18 |
| 2. | .4.15 | Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level | 18 |
| 2. | .4.16 | Changes in Laboratory Test Values (Glucose Metabolism) | 18 |
| 2. | .4.17 | Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications> | 19 |
| 2. | .4.18 | Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications > | 19 |
| 2.5 | Effic | cacy Statistical Analysis | 20 |
| 2. | .5.1 | Changes in Laboratory Test Values (Fasting Lipid) | 20 |
| 2. | .5.2 | Changes in Laboratory Test Values (Random Lipid) | 20 |
| | 2.5.3 | Changes in Fasting Lipid-Related Ratio. | 20 |
|---|---|---|---|
| | 2.5.4 | Changes in Fasting Triglyceride by Factor of Patient Demographics and Treatment Details | 21 |
| | 2.5.5 | Changes in Random Triglyceride by Factor of Patient Demographics and Treatment Details | 22 |
| 3.0 | .0 Summary of Onset Status of Serious Adverse Events (Exhibit 2-2) | | 23 |

#### 1.0 Definitions of Terms

# 1.1 Definitions

| Item | Definition |
|---|---|
| Survey unit period | Periodic Safety Report 1: July 22, 2012 to January 21, 2013 |
| (periodic safety report) | Periodic Safety Report 2: January 22, 2013 to July 21, 2013 |
| | Periodic Safety Report 3: July 22, 2013 to January 21, 2014 |
| | Periodic Safety Report 4: January 22, 2014 to July 21, 2014 |
| | Periodic Safety Report 5: July 22, 2014 to July 21, 2015 |
| | Periodic Safety Report 6: July 22, 2015 to July 21, 2016 |
| | Periodic Safety Report 7: July 22, 2016 to July 21, 2017 |
| Drug | Lotriga Granular Capsules |
| SOC | System organ class of MedDRA. |
| HLGT | High level group term of MedDRA. |
| PT | Preferred term of MedDRA. |
| LLT | Lowest level term of MedDRA. |
| Enrolled patient | A patient approved for enrollment in the Study. |
| Patient with eCRF | An enrolled patient whose eCRF was submitted via |
| collected | |
| Patient with eCRF | An enrolled patient other than a patient with eCRF collected. |
| uncollected | |
| Locked patient | A patient who has completed the approval process in the PMS system. |
| Unlocked patient | A patient with eCRF collected other than a locked patient. |
| Safety-evaluable patient | A locked patient included in safety evaluation. |
| Safety-unevaluable patient | A locked patient excluded from safety evaluation. |
| Efficacy-evaluable patient | A safety-evaluable patient included in efficacy evaluation. |
| Efficacy-unevaluable | A safety-evaluable patient excluded from efficacy evaluation. |
| patient | |
| ADR | An abbreviated form of the term 'adverse drug reaction or infection.' |
| | Refers to an adverse event other than those judged by the investigator as 'not |
| | related' in causality to the Drug. |
| | In this plan, 'adverse drug reactions or infections' is used in headings, and |
| | 'ADRs' is used in the text and tables. |
| Serious adverse event | [Prior-approval data] |
| (SAE) | An adverse event (AE) judged as 'serious' by the trial investigator. |
| | [Surveillance data] |
| | An adverse event (AE) judged as 'serious' by the investigator. |
| | Note that events listed in the separate MedDRA code list of the Takeda |
| | Medically Significant AE List should be treated as serious even if judged as |
| | 'not serious' by the investigator. |

| Item | Definition |
|---|---|
| Bleeding-related event | An event falling under Standardized MedDRA Query (SMQ) code 20000038 |
| | (hemorrhagic SMQ [narrow scope]). |
| Rate of patients | [For safety compilation with safety-evaluable patients] |
| | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Evaluable Patients] × 100. |
| | [For safety compilation with safety-unevaluable patients] |
| | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Unevaluable Patients] × 100. |
| Incidence | [For safety compilation with safety-evaluable patients] |
| | Calculated by the following equation: [Number of Events] / [Number of |
| | Safety-Evaluable Patients] × 100. |
| | [For safety compilation with safety-unevaluable patients] |
| | Calculated by the following equation: [Number of Events] / [Number of |
| | Safety-Unevaluable Patients] × 100. |
| Onset time | Calculated by the following equation: [Onset Date] - [Start Date] + 1. |
| | If the onset date is unknown, use the first day of the month instead in this |
| | equation. However, use the start date if [Start Year & Month] = [Onset Year & |
| | Month]. |
| Liver patient | A patient with 'fatty liver,' 'alcoholic fatty liver,' 'chronic hepatitis' or 'hepatic |
| | cirrhosis' check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SMQ code 20000005 (hepatic SMQ [narrow |
| | scope]) in the Complication Details (Other Diseases) field. |
| Kidney patient | A patient with 'diabetic nephropathy,' 'glomerulonephritis' or 'chronic kidney |
| | disease (CKD)' check-marked in the Complication Details field. Or a patient |
| | with a complication falling under the Takeda MedDRA query (TMQ) (Renal |
| | Disease) in the Complication Details (Other Diseases) field. |
| Heart patient | A patient with 'myocardial infarction,' 'angina pectoris' or 'atrial fibrillation' |
| | check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SOC code 10007541 (cardiac disorders) in the |
| | Complication Details (Other Diseases) field. |
| Cerebrovascular patient | A patient with 'cerebral infarction' or 'cerebral hemorrhage' check-marked in |
| | the Complication Details field. Or a patient with a complication falling under |
| | the SMQ code 20000060 (cerebrovascular SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Diabetic patient | A patient with 'diabetes' check-marked in the Complication Details field. Or a |
| | patient with a complication falling under the TMQ code (Diabetes Mellitus |
| | Confirmed diagnosis, excl diagnostics) in the Complication Details (Other |
| | Diseases) field. |

| Item | Definition |
|---|---|
| Hypertensive patient | A patient with 'hypertension' check-marked in the Complication Details field. |
| | Or a patient with a complication falling under the SMQ code 20000147 |
| | (hypertensive SMQ [narrow scope]) in the Complication Details (Other |
| | Diseases) field. |
| Myocardial infarction | A patient with 'myocardial infarction' check-marked in the Complication |
| patient | Details field. Or a patient with a complication falling under the SMQ code |
| | 20000047 (myocardial infarction SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Anginal patient | A patient with 'angina pectoris' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10002383 (angina pectoris), 10002388 (unstable angina pectoris), 10036759 |
| | (Prinzmetal angina), or 10058144 (postinfarction angina) in the Complication |
| | Details (Other Diseases) field. |
| Atrial fibrillation patient | A patient with 'atrial fibrillation' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10003658 (atrial fibrillation) in the Complication Details (Other Diseases) |
| | field. |
| Ischemic cerebrovascular | A patient with 'cerebral infarction' check-marked in the Complication Details |
| patient | field. Or a patient with a complication falling under the SMQ code 20000063 |
| | (ischemic cerebrovascular disease SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Hemorrhagic | A patient with 'cerebral hemorrhage' check-marked in the Complication Details |
| cerebrovascular patient | field. Or a patient with a complication falling under the SMQ code 20000064 |
| | (hemorrhagic cerebrovascular disease SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Bleeding-related event | A patient with a complication falling under the SMQ code 20000038 (bleeding |
| patient | SMQ [narrow scope]) in the Complication Details (Other Diseases) field. |
| Age | Calculated by the following equation: [Start Year] - [Birth Year] - 1 if [Start |
| | Month & Day] < [Birth Month & Day]. |
| | Calculated by the following equation: [Start Year] - [Birth Year] if [Start Month |
| | & Day] ≥ [Birth Month & Day]. |
| | If the birth day is unknown, use the first day of the month instead in this |
| | equation. |
| BMI | Calculated by the following equation: [Weight (kg)] / (0.0001 × [Height (cm)] |
| | × [Height (cm)]). Indicated by rounding off to the first decimal place. |
| Disease duration (in years) | Calculated by the following equation: ([Start Year & Month] - [Year & Month] |
| | of Hyperlipidemia Diagnosis] + 1) / 12. Indicated by rounding off to the first |
| | decimal place. |

| Item | Definition |
|---|---|
| Start date | The start date of first administration of the Drug stated in the Treatment |
| | Duration field of the eCRF. |
| End date | The end date of last administration of the Drug stated in the Treatment Duration |
| | field of the eCRF. |
| | However, if the end date of last administration is in 'ongoing 12 months after |
| | baseline,' the end date should be the start date plus 360 days. |
| Observation period (in | Calculated by the following equation: [End Date] - [Start Date] + 1. |
| days) | |
| Treatment duration (in | A total of ([End Date] - [Start Date] + 1) in the number of actual administration |
| days) | days, excluding washout period. |
| Mean daily dose | Calculated by the following equation: Total of ([Daily Dose] × [Total Period of |
| | Treatment with the Dose]) / [Observation Period]. See the above for calculation |
| | of observation period. |
| Concomitant medication | A drug used during the surveillance period. However, concomitant medications |
| | exclude drugs used for adverse events occurring during the period. |
| Antihyperlipidemic drug | A drug starting with any of the following drug codes: 218, 2190006, 2190101, |
| | 2190102, 2190103, 2190104, 290006, 3133001, 3133400, 3399004. |
| Statins drug | A drug starting with any of the following drug codes: 2189010, 2189011, |
| | 2189012, 2189015, 2189016, 2189017. |
| Fibrate drug | A drug starting with drug code: 2183. |
| Intestinal transporter | A drug starting with drug code: 2189018. |
| inhibitor | |
| Anion-exchange resin | A drug starting with any of the following drug codes: 2189009, 2189014. |
| Nicotinic acid derivative | A drug starting with any of the following drug codes: 2189004, 2189005, |
| | 2190006. |
| Probucol | A drug starting with drug code: 2189008. |
| Ethyl icosapentate (EPA) | A drug starting with drug code: 3399004. |
| Anticoagulant drug | A drug starting with any of the following drug codes: 333, 2190408, 6343424. |
| Antiplatelet drug | A drug starting with any of the following drug codes: 3399 (excluding |
| | 3399004), 2171010, 2171402. |
| Anticoagulant/antiplatelet | A drug that falls under the class of either anticoagulant or antiplatelet drugs |
| drug | |
| LDL cholesterol | Calculated the equation below if the patient is fasting at the time of blood |
| (Friedewald formula) | collection for laboratory testing with triglyceride 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol - triglyceride / 5 |
| Non-HDL cholesterol | Calculated by the equation below if triglyceride is 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |

| Item | Definition |
|---|---|
| | Total cholesterol - HDL cholesterol |
| TC/LDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | Total cholesterol / LDL cholesterol (Friedewald formula) |
| LDL-C/HDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / HDL cholesterol |
| LDL-C/Apo-B ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / Apo-B |
| Summary statistics | Mean value, standard deviation, minimum value, first quartile, median, third |
| | quartile, maximum value |

#### 1.2 Number of Display Digits

| Item | Definition |
|---|---|
| Percentage (%) Rate of patients with ADRs: | |
| | Indicated by rounding off to the second decimal place. |
| | Other than above: |
| | Indicated by rounding off to the first decimal place. |
| Summary statistics | Mean value: |
| | Indicated by rounding off to the first digit below the raw numerical data. |
| | Standard deviation: |
| | Indicated by rounding off to the second digit below the raw numerical data. |
| | First quartile, median, third quartile: |
| | Indicated by rounding off to the first digit below the raw numerical data. |
| | Minimum value, maximum value: |
| | Indicated at the same digits of the raw numerical data. |
| Confidence interval | Indicated by rounding off to the second digit below the raw numerical data. |
| p value | Indicated by rounding down to the third decimal place. |
| | Expressed as p<0.001 when rounding down at the forth decimal place makes the |
| | figure below 0.001. |

#### 1.3 Level of Significance

Two-sided 5%

#### 1.4 Handling of Evaluation Timepoint Data

The evaluation timepoints are the start of treatment with the Drug (baseline), Month 3, Month 6, Month 9, Month 12, and final evaluation timepoint.

If multiple data exist within each evaluation timepoint, calculate absolute values of difference in measurement intervals from the basic day count and adopt the minimum absolute value as date for that evaluation timepoint. If all the absolute values are the same, adopt one for the latest date of testing/measurement. Test/Measurement values should not be adopted that have been obtained after completion of treatment with the Drug. The final evaluation timepoint test/measurement should be one taken on the latest date within 405 days elapsed since the start date (including values tested/measured during washout period). Note that the number days elapsed since the start date should be counted with the start date as day 0 and the previous day as day -1.

| Evaluation Timepoint | Tolerance<br>(Number of Days Since Baseline) | Basic Day Count |
|---|---|---|
| Baseline | -90 to 0 | 0 |
| Month 3 | 1 to 135 | 90 |
| Month 6 | 136 to 225 | 180 |
| Month 9 | 226 to 315 | 270 |
| Month 12 | 316 to 405 | 360 |
| Final evaluation | 1 to 405 | - |
| timepoint | | |

#### 2.0 Results of Special Drug Use Surveillance (Survey 1)

<Lotriga Granular Capsules Special Drug Use Surveillance [long-term use survey]>

#### 2.1 Patient Breakdown (Patient Disposition)

| Statistical Analysis | Enrolled patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Number of enrolled patients, number of patient enrollment sites, number of patients |
| Statistical Analysis | with eCRFs collected, number of patients with eCRFs uncollected, number of locked |
| | patients, number of unlocked patients, number of safety-evaluable patients, number |
| | safety-unevaluable patients, number of efficacy-evaluable patients, number |
| | efficacy-unevaluable patients |
| | Do not double-count the same medical institution with different participating clini |
| | departments when counting the number of patient enrollment sites. |
| | Count the number of patients per reason below for not collecting and total the |
| | numbers when the number of patients with eCRFs uncollected. |
| | <reasons collecting="" for="" not=""></reasons> |
| | Survey under way |
| | eCRFs uncollectable |
| | Investigator transferred |
| | • Investigator's health reasons |
| | • Patients enrolled 15 days after Drug prescription [before eCRF collection] |
| | • Others |
| | Count the number of patients per reason below for exclusion and total the numbers |
| | when counting the numbers of safety- and efficacy-unevaluable patients. If the same |
| | patient falls under multiple reasons for exclusion, they should be counted separately. |
| | <reasons evaluation="" exclusion="" for="" from="" safety=""></reasons> |
| | Drug administered before contract period |
| | Patient enrolled 15 days after Drug prescription |
| | No data available after Drug administration |
| | Drug not administered |
| | <reasons efficacy="" evaluation="" exclusion="" for="" from=""></reasons> |
| | Pre- or post-administration lipid-related values (fasting or random) unavailable |
| | No output needs to be generated for items for which the number of patients is zero. |
| | For periodic safety reports, the numbers of efficacy-evaluable and unevaluable |
| | patients should not be counted. |
| Figure/Table No. | Figure 2.1, Table 2.1 |

#### 2.2 Patient Demographics

| Statistical Analysis Set | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Details of | | |
| Statistical Analysis | compile the number of patients and incidence. Item Name Category | |
| | Sex | Male, Female |
| | Age | Summary statistics |
| | | Minimum age to 64 years, 65 to 74 years, 75 years to |
| | | maximum age, Unknown |
| | Treatment category | Outpatient, inpatient |
| | BMI | Summary statistics |
| | | Less than $18.5 \text{ kg/m}^2$ , $18.5 \text{ to less than } 25 \text{ kg/m}^2$ , $25 \text{ to}$ |
| | | less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | | Hypertension, Diabetic, Liver disorder, Kidney |
| | | disorder, Cardiac disorders [myocardial infarction, |
| | Complication | angina pectoris, atrial fibrillation, others], |
| | breakdown | Cerebrovascular diseases [hemorrhagic |
| | | cerebrovascular disease, ischemic cerebrovascular |
| | | disease, others], Bleeding-related event, Others |
| | Drinking history | |
| | (Does the patient | |
| | drink alcoholic | Yes, No, Unknown |
| | beverages nearly | |
| | every day?) | T d 150 /H 150 / H 400 /H 400 |
| | | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | Fraincasial contact | to less than 500 mg/dL, 500mg/dL or over, Not measured |
| | Fasting triglyceride at | |
| | baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | | 750 mg/dL or over, Not measured |
| | | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | | to less than 500 mg/dL, 500mg/dL or over, Not |
| | Random triglyceride | measured |
| | at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 |
| | | to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | | 750 mg/dL or over, Not measured |

| | Smoking history | Never, Current, Former, Unknown |
|---|---|---|
| | Hypersensitivity disposition | No, Yes, Unknown |
| | | Summary statistics |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence of surgery within one month before baseline | No, Yes |
| | Pregnancy status during treatment (only for female) | No, Yes |
| Figure/Table No. | Table 2.2 | |

#### 2.3 Treatment Details

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize the patient population by the following categories for each item and | |
| Statistical Analysis | compile the number of patients and incidence. | |
| | Item Name | Category |
| | Initial dose | 2 g, 4 g, Other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) | No, Yes |
| | Breakdown of concomitant medications (during observation period) | Antihyperlipidemic drugs [statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others], Anticoagulant/antiplatelet drugs [anticoagulant drugs, antiplatelet drugs] |
| | Completion of treatment with the Drug | No, Yes, Unknown |
| | Reason for treatment completion | Treatment goal achieved, AE developing, Patient no longer visiting hospital due to hospital transfer or otherwise, Insufficient effect, Other |
| Figure/Table No. | Table 2.3 | |

### 2.4 Safety Statistical Analysis

#### 2.4.1 Onset Status of Adverse Drug Reactions or Infections (Exhibit 2)

| Statistical Analysis | Safety-evaluable natients in | clinical studies before approval (total of natients in |
|---|---|---|
| Set | Safety-evaluable patients in clinical studies before approval (total of patients in | |
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the | |
| | Adverse Drug Reactions section of the package insert) and this special drug use | |
| | surveillance | |
| Details of | Compile the following items for the prior-approval status and per survey unit period | |
| Statistical Analysis | of the special drug use surveil | |
| | Statistical analysis of 'number | r of study sites,' 'number of surveyed patients,' 'number |
| | of patients with ADRs,' and 'r | number of ADRs' should cover safety-evaluable patients |
| | locked during each survey uni | |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients with ADRs | Number of patients in which ADRs occurred. |
| | Number of ADRs | Number of ADRs that occurred. Every PT occurring should be counted as one event. |
| | Rate of patients with ADRs | Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Evaluable Patients] × 100 |
| | ADR type | Categorize by SOC and compile ADRs by PT in each category. In the case of laboratory testing, categorize by SOC, summarize by HLGT, and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. At PT level, the numbers of ADRs should be presented by PT code in ascending order. If adverse drug reactions (LLTs) under the same PT occur more than once in the same patient, they should be counted as one PT. |
| | Cumulative total for special drug use surveillance | A respective total of the numbers of study sites and patients per survey unit period. Do not double-count the same medical institution when counting the number of study sites. |
| Figure/Table No. | Table 2.4.1 | |

#### 2.4.2 Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients

| Statistical Analysis | Safety-unevaluable patients in clinical studies before approval (total of patients in | |
|---|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the | |
| | Adverse Drug Reactions section of the package insert) and this specified drug use | |
| | surveillance | |
| Details of | Compile the following items. | |
| Statistical Analysis | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-unevaluable patients. |
| | Number of patients with ADRs | Number of patients in which ADRs occurred. |
| | Number of ADRs | Number of ADRs that have occurred. Every PT occurring should be counted as one event. |
| | Rate of patients with ADRs | Calculated by the following equation: [Number of Patients with ADRs] / [Number of Safety-Unevaluable Patients] × 100 |
| | ADR type | Categorize by SOC and compile ADRs by PT in each category. In the case of laboratory testing, categorize by SOC, summarize by HLGT, and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. At PT level, the numbers of ADRs should be presented by PT code in ascending order. If adverse drug reactions (LLTs) under the same PT occur more than once in the same patient, they should be counted as one PT. |
| Figure/Table No. | Table 2.4.2 | |

#### 2.4.3 Onset Status of AE

| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in |
|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the |
| | Adverse Drug Reactions section of the package insert) and this special drug use |
| | surveillance |
| Details of | The compilation method is the same as described in section 2.4.1. However, adverse |
| Statistical Analysis | drug reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.3 |

#### 2.4.4 Onset Status of Adverse Events in Safety-Unevaluable Patients

| Statistical Analysis | Safety-unevaluable patients in clinical studies before approval (total of patients in |
|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the |
| | Adverse Drug Reactions section of the package insert) and this specified drug use |
| | surveillance |
| Details of | Compilation method is the same as described in section 2.4.2. However, adverse drug |
| Statistical Analysis | reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.4 |

#### 2.4.5 Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADRs by the following categories for each item and compile ADR types. | |
| Statistical Analysis | Item Name | Details of Statistical Analysis |
| | Number of patients | Compile the number of patients with ADRs. |
| | Number of ADRs | At SOC, the number of ADRs should be compiled by totaling associated PTs that occurred. At PT level, every PT occurring should be counted as one event. |
| | Item Name | Category |
| | Seriousness | Serious, Not serious |
| | Onset time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over, Unknown |
| | Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, Death, Unknown |
| Figure/Table No. | Table 2.4.5 | |

#### 2.4.6 Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize AEs by the following categories for each item and compile AE types. | |
| Statistical Analysis | The compilation method of AE types is the same as described in section 2.4.5. | |
| | However, adver | rse drug reactions should be replaced by adverse events. |
| | Item Name | Category |
| | Seriousness | Serious, Not serious |
| | Ongot time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to |
| | Onset time | 360 days, 361 days or over, Unknown |
| | Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, |
| | Outcome | Death, Unknown |
| | Causal | Related, Not related, Unevaluable |
| | relationship | If AEs (LLTs) occur more than once in the same patient, they |
| | with the | should be counted as one event in the following order of priority: |
| | Drug | (1) Related, (2) Unevaluable, (3) Not related |
| Figure/Table No. | Table 2.4.6 | |

# 2.4.7 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Time,

and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Categorize adverse drug reactions (bleeding-related events) by the following |
| Statistical Analysis | categories for each item, and count the types of adverse drug reactions |
| | (bleeding-related events). |
| | The categories and the compilation method of adverse drug reactions are the same as |
| | described in section 2.4.5. |
| Figure/Table No. | Table 2.4.7 |

# 2.4.8 Rate of Patients of Adverse Drug Reactions or Infections by Factor of Patient Demographics andTreatment Details

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADRs by the following categories for each item and compile the rate of | |
| Statistical Analysis | patients with ADRs (point estimate and 95% confidence interval). | |
| | Perform Fisher's exact test for items having categories without rank order, and | |
| | - | items having categories with rank order. |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to |
| | | maximum age, Unknown |
| | BMI | Less than $18.5 \text{ kg/m}^2$ , $18.5 \text{ to less than } 25 \text{ kg/m}^2$ , $25 \text{ to }$ |
| | DIVII | less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | | Hypertension, Diabetic, Liver disorder, Kidney |
| | | disorder, Cardiac disorders [myocardial infarction, |
| | Complication | angina pectoris, atrial fibrillation, others], |
| | breakdown | Cerebrovascular diseases [hemorrhagic |
| | | cerebrovascular disease, ischaemic cerebrovascular |
| | | disease, others], Bleeding-related event, Others |
| | Drinking history | |
| | (Does the patient | |
| | drink alcoholic | Yes, No, Unknown |
| | beverages nearly | |
| | every day?) | |
| | | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | | to less than 500 mg/dL, 500mg/dL or over, Not |
| | Fasting triglyceride at | measured |
| | baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 |
| | | to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | | 750 mg/dL or over, Not measured |
| | Random triglyceride | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured |
| | at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |

| | Smoking history | Never, Current, Former, Unknown |
|---|---|---|
| | Hypersensitivity disposition | No, Yes, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence of surgery within one month before baseline | No, Yes |
| | Pregnancy status during treatment (only for female) | No, Yes |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) | No, Yes |
| | Breakdown of concomitant medications (during observation period) | Antihyperlipidemic drugs [statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others], Anticoagulant/antiplatelet drugs [anticoagulant drugs, antiplatelet drugs] |
| Figure/Table No. | Table 2.4.8 | |

#### 2.4.9 Onset Status of Adverse Drug Reactions or Infections by Age Group

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Classify the patient population into 64 years or below, 65 to 74 years, and 75 years or |
| Statistical Analysis | over, and compile ADR types. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.9 |

#### 2.4.10 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Liver

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of liver complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.10 |

#### 2.4.11 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kidney

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of kidney complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.11 |

## 2.4.12 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant

#### Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant anticoagulant and/or |
| Statistical Analysis | antiplatelet drugs (Both, Anticoagulant only, Antiplatelet only, Neither). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.12 |

# 2.4.13 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence of Concomitant Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile the types of adverse drug reactions (bleeding-related events) by presence or |
| Statistical Analysis | absence of concomitant anticoagulant and/or antiplatelet drugs (Both, Anticoagulant |
| | only, Antiplatelet only, Neither). |
| | The compilation method of the types of adverse drug reactions is the same as |
| | described in section 2.4.1. |
| Figure/Table No. | Table 2.4.13 |

#### 2.4.14 Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose fasting |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline fasting triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 $$ |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.14 |

#### 2.4.15 Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose random |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline random triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 $$ |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.15 |

#### 2.4.16 Changes in Laboratory Test Values (Glucose Metabolism)

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseli |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. Also perform the corresponding t-test. |
| Figure/Table No. | Table 2.4.16 |

#### 2.4.17 Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. Also perform the corresponding t-test. |
| Remarks | Stratification factor: With diabetic complications |
| Figure/Table No. | Table 2.4.17 |

#### 2.4.18 Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. Also perform the corresponding t-test. |
| Remarks | Stratification factor: Without diabetic complications |
| Figure/Table No. | Table 2.4.18 |

#### 2.5 Efficacy Statistical Analysis

#### 2.5.1 Changes in Laboratory Test Values (Fasting Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), total cholesterol |
| | (mg/dL), LDL cholesterol (direct measurement) (mg/dL), LDL cholesterol |
| | (Friedewald formula) (mg/dL), HDL cholesterol (mg/dL), non-HDL cholesterol |
| | (mg/dL), VLDL cholesterol (mg/dL), Apo-AI (mg/dL), Apo-B (mg/dL), Apo-CIII |
| | (mg/dL), lipoprotein(a) (mg/dL), and remnant lipoprotein cholesterol (mg/dL). In |
| | addition, calculate the 95% confidence interval for the mean value for rates of change |
| | from baseline (%). Also perform the corresponding t-test. |
| Figure/Table No. | Table 2.5.1 |

#### 2.5.2 Changes in Laboratory Test Values (Random Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom random |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for random measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), total cholesterol |
| | (mg/dL), LDL cholesterol (direct measurement) (mg/dL), HDL cholesterol (mg/dL), |
| | non-HDL cholesterol (mg/dL), VLDL cholesterol, Apo-AI (mg/dL), Apo-B (mg/dL), |
| | Apo-CIII (mg/dL), lipoprotein(a) (mg/dL), and remnant lipoprotein cholesterol |
| | (mg/dL). In addition, calculate the 95% confidence interval for the mean value for |
| | rates of change from baseline (%). Also perform the corresponding t-test. |
| Figure/Table No. | Table 2.5.2 |

#### 2.5.3 Changes in Fasting Lipid-Related Ratio

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for TC/LDL-C, |
| Statistical Analysis | LDL-C/HDL-C, and LDL-C/Apo-B. |
| Figure/Table No. | Table 2.5.3 |

#### 2.5.4 Changes in Fasting Triglyceride by Factor of Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting | |
|---|---|---|
| Set | blood collection was performed at baseline | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of fasting | |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | ВМІ | Less than 18.5kg/m <sup>2</sup> , 18.5 to less than 25kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Fasting triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) (antihyperlipidemic drugs) | No, Yes |
| | Breakdown of concomitant medications (during observation period) (antihyperlipidemic drugs) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |
| Figure/Table No. | Figure/Table No. Table 2.5.4 | |

#### 2.5.5 Changes in Random Triglyceride by Factor of Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom random | |
|---|---|---|
| Set | blood collection was performed at baseline | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of random | |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | BMI | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) (antihyperlipidemic drugs) | No, Yes |
| | Breakdown of concomitant medications (during observation period) (antihyperlipidemic drugs) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |
| Figure/Table No. | Table 2.5.5 | |

#### 3.0 Summary of Onset Status of Serious Adverse Events (Exhibit 2-2)

| Statistical Analysis | | |
|---|---|---|
| Set | linical studies inside and outside Japan used for safety evaluation stated in the | |
| | Adverse Drug Reactions section of the package insert) and this special drug use | |
| Details of | surveillance Compile the following items per survey unit period of the prior-approval status and of | |
| Statistical Analysis | | ne special drug use surveillance. |
| Statistical Alialysis | | nber of study sites,' 'number of surveyed patients,' 'number |
| | of patients,' and 'number | of SAEs' should cover safety-evaluable patients locked |
| | during each survey unit pe | |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients | Number of patients with SAEs |
| | Number of SAEs | Number of SAEs Every PT occurring should be counted as one event. |
| | Rate of patients | Calculated by the following equation: [Number of Patients with SAEs] / [Number of Safety-Evaluable Patients] × 100. |
| | SAE type | Categorize by SOC and compile ADRs by PT in each category. In the case of laboratory testing, categorize by SOC, summarize by HLGT, and compile ADRs by PT. At SOC level, the numbers and rates of patients with SAEs should be presented by SOC internationally agreed order. At PT level, the numbers of SAEs should be presented by PT code in ascending order. If SAEs (LLTs) under the same PT occur more than once in the same patient, they should be counted as one PT. The number of SAEs of which causal relationship to the Drug has been denied should be entered in the [ ] brackets. |
| | Cumulative total of special drug use surveillance | patients per survey unit period. |
| Figure/Table No. | Table 3.0 | |

## Statistical Analysis Plan

# (for Periodic Safety Reporting/Reexamination Application) <Lotriga Granular Capsules>

Takeda Pharmaceutical Company Limited

Pharmacovigilance Department, Pharmaceutical Development Division
Postmarketing Surveillance Group Manager

PPD

Statistical Analysis Contractor

PPD

#### Table of Contents

| 1.0 | Defini | tions of Terms | 1 |
|---|---|---|---|
| 1.1 | Def | initions | 1 |
| 1.2 | Nur | nber of Display Digits | 5 |
| 1.3 | Lev | el of Significance | 5 |
| 1.4 | Har | ndling of Evaluation Timepoint Data | 6 |
| 2.0 | Result | s of Special Drug Use Surveillance (Survey 1) | 7 |
| 2.1 | Pati | ent Breakdown (Patient Disposition) | 7 |
| 2.2 | Pati | ent Demographics | 7 |
| 2.3 | Trea | atment Details | 10 |
| 2.4 | Safe | ety Statistical Analysis | .11 |
| 2. | 4.1 | Onset Status of Adverse Drug Reactions or Infections (Exhibit 2) | .11 |
| 2. | 4.2 | Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients (Exhibit 2) | 12 |
| 2. | 4.3 | Onset Status of AE | 13 |
| 2. | 4.4 | Onset Status of Adverse Events in Safety-Unevaluable Patients | 13 |
| 2. | 4.5 | Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome | 13 |
| 2. | 4.6 | Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome | 14 |
| 2. | 4.7 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Tire | ne, |
| ar | nd Outo | come | 14 |
| 2. | 4.8 | Rate of Patients of Adverse Drug Reactions or Infections by Factor of Patient Demographics a | ınd |
| Ti | reatmei | nt Details | 15 |
| 2. | 4.9 | Onset Status of Adverse Drug Reactions or Infections by Age Group | 17 |
| 2. | 4.10 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Live | ver |
| C | omplic | ations | 17 |
| 2. | 4.11 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kidr | ıey |
| C | omplic | ations | 17 |
| 2. | 4.12 | Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomita | ant |
| A | nticoag | gulant and/or Antiplatelet Drugs | |
| | 4.13 | Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence | |
| C | oncom | itant Anticoagulant and/or Antiplatelet Drugs | |
| 2. | 4.14 | Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level | 18 |
| 2. | 4.15 | Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level | |
| 2. | 4.16 | Changes in Laboratory Test Values (Glucose Metabolism) | 19 |
| | 4.17 | Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications > | |
| | 4.18 | Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications > | |
| 2.5 | | cacy Statistical Analysis | |
| | 5.1 | Changes in Laboratory Test Values (Fasting Lipid) | |
| 2 | 5.2 | Changes in Laboratory Test Values (Random Lipid) | 20 |

| | 2.5.3 | Changes in Fasting Lipid-Related Ratio. | . 20 |
|---|---|---|---|
| | 2.5.4 | Changes in Fasting Triglyceride by Factor of Patient Demographics and Treatment Details | . 21 |
| | 2.5.5 | Changes in Random Triglyceride by Factor of Patient Demographics and Treatment Details | . 22 |
| 3.0 | Summa | ary of Onset Status of Serious Adverse Events (Exhibit 2-2) | . 23 |

#### 1.0 Definitions of Terms

# 1.1 Definitions

| Item | Definition |
|---|---|
| Survey unit period | Periodic Safety Report 3: July 22, 2013 to January 21, 2014 |
| (periodic safety report) | Periodic Safety Report 4: January 22, 2014 to July 21, 2014 |
| | Periodic Safety Report 5: July 22, 2014 to July 21, 2015 |
| | Periodic Safety Report 6: July 22, 2015 to July 21, 2016 |
| | Periodic Safety Report 7: July 22, 2016 to July 21, 2017 |
| Drug | Lotriga Granular Capsules |
| SOC | System organ class of MedDRA. |
| HLGT | High level group term of MedDRA. |
| PT | Preferred term of MedDRA. |
| LLT | Lowest level term of MedDRA. |
| Enrolled patient | A patient approved for enrollment in the Study. |
| Patient with eCRF | A patient finalized in CCI. |
| collected | |
| Patient with eCRF | An enrolled patient other than a patient with eCRF collected. |
| uncollected | |
| Locked patient | A patient who has completed the approval process in the PMS system. |
| Unlocked patient | A patient with eCRF collected other than a locked patient. |
| Safety-evaluable patient | A patient listed as 'evaluable' for safety in the evaluability sheet. |
| Safety-unevaluable patient | A patient listed as 'unevaluable' for safety in the evaluability sheet. |
| Efficacy-evaluable patient | A safety-evaluable patient listed as 'evaluable' for efficacy in the evaluability |
| | sheet. |
| Efficacy-unevaluable | A safety-evaluable patient listed as 'unevaluable' for efficacy in the evaluability |
| patient | sheet. |
| ADR | An abbreviated form of the term 'adverse drug reaction or infection.' |
| | Refers to an adverse event other than those judged by the investigator as 'not |
| | related' in causality to the Drug. |
| | In this plan, 'adverse drug reactions or infections' is used in headings, and |
| | 'ADRs' is used in the text and tables. |
| Serious adverse event | An adverse event (AE) judged as 'serious' by the investigator. |
| (SAE) | Note that events listed in the separate MedDRA code list of the Takeda |
| | Medically Significant AE List should be treated as serious even if judged as |
| | 'not serious' by the investigator. |
| Bleeding-related event | An event falling under Standardized MedDRA Query (SMQ) code 20000038 |
| | (hemorrhagic SMQ [narrow scope]). |
| Rate of patients | Calculated by the following equation: [Number of Patients] / [Number of |
| | Safety-Evaluable Patients] × 100. |

| Item | Definition |
|---|---|
| Incidence | Calculated by the following equation: [Number of Events] / [Number of |
| | Safety-Evaluable Patients] × 100. |
| Onset time | Calculated by the following equation: [Onset Date] - [Start Date] + 1. |
| | If the onset date is unknown, use the first day of the month instead in this |
| | equation. However, use the start date if [Start Year & Month] = [Onset Year & |
| | Month]. |
| Liver patient | A patient with 'fatty liver,' 'alcoholic fatty liver,' 'chronic hepatitis' or 'hepatic |
| | cirrhosis' check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SMQ code 20000005 (hepatic SMQ [narrow |
| | scope]) in the Complication Details (Other Diseases) field. |
| Kidney patient | A patient with 'diabetic nephropathy,' 'glomerulonephritis' or 'chronic kidney |
| | disease (CKD)' check-marked in the Complication Details field. Or a patient |
| | with a complication falling under the Takeda MedDRA query (TMQ) (Renal |
| | Disease) in the Complication Details (Other Diseases) field. |
| Heart patient | A patient with 'myocardial infarction,' 'angina pectoris' or 'atrial fibrillation' |
| | check-marked in the Complication Details field. Or a patient with a |
| | complication falling under the SOC code 10007541 (cardiac disorders) in the |
| | Complication Details (Other Diseases) field. |
| Cerebrovascular patient | A patient with 'cerebral infarction' or 'cerebral hemorrhage' check-marked in |
| | the Complication Details field. Or a patient with a complication falling under |
| | the SMQ code 20000060 (cerebrovascular SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Diabetic patient | A patient with 'diabetes' check-marked in the Complication Details field. Or a |
| | patient with a complication falling under the TMQ code (Diabetes Mellitus |
| | Confirmed diagnosis, excl diagnostics) in the Complication Details (Other |
| | Diseases) field. |
| Hypertensive patient | A patient with 'hypertension' check-marked in the Complication Details field. |
| | Or a patient with a complication falling under the SMQ code 20000147 |
| | (hypertensive SMQ [narrow scope]) in the Complication Details (Other |
| | Diseases) field. |
| Myocardial infarction | A patient with 'myocardial infarction' check-marked in the Complication |
| patient | Details field. Or a patient with a complication falling under the SMQ code |
| | 20000047 (myocardial infarction SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Anginal patient | A patient with 'angina pectoris' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10002383 (angina pectoris), 10002388 (unstable angina pectoris), 10036759 |
| | (Prinzmetal angina), or 10058144 (postinfarction angina) in the Complication |

| Item | Definition |
|---|---|
| | Details (Other Diseases) field. |
| Atrial fibrillation patient | A patient with 'atrial fibrillation' check-marked in the Complication Details |
| | field. Or a patient with a complication falling under the MedDRA PT code |
| | 10003658 (atrial fibrillation) in the Complication Details (Other Diseases) |
| | field. |
| Ischemic cerebrovascular | A patient with 'cerebral infarction' check-marked in the Complication Details |
| patient | field. Or a patient with a complication falling under the SMQ code 20000063 |
| | (ischemic cerebrovascular disease SMQ [narrow scope]) in the Complication |
| | Details (Other Diseases) field. |
| Hemorrhagic | A patient with 'cerebral hemorrhage' check-marked in the Complication Details |
| cerebrovascular patient | field. Or a patient with a complication falling under the SMQ code 20000064 |
| | (hemorrhagic cerebrovascular disease SMQ [narrow scope]) in the |
| | Complication Details (Other Diseases) field. |
| Age | Calculated by the following equation: [Start Year] - [Birth Year] - 1 if [Start |
| | Month & Day] < [Birth Month & Day]. |
| | Calculated by the following equation: [Start Year] - [Birth Year] if [Start Month |
| | & Day] ≥ [Birth Month & Day]. |
| | If the birth day is unknown, use the first day of the month instead in this |
| | equation. |
| BMI | Calculated by the following equation: [Weight (kg)] / (0.0001 × [Height (cm)] |
| | × [Height (cm)]). Indicated by rounding off to the first decimal place. |
| Disease duration (in years) | Calculated by the following equation: ([Start Year & Month] - [Year & Month] |
| | of Hyperlipidemia Diagnosis] + 1) / 12. Indicated by rounding off to the first |
| | decimal place. |
| Start date | The start date of first administration of the Drug stated in the Treatment |
| | Duration field of the eCRF. |
| End date | The end date of last administration of the Drug stated in the Treatment Duration |
| | field of the eCRF. |
| | However, if the end date of last administration is in 'ongoing 12 months after |
| | baseline,' the end date should be the start date plus 360 days. |
| Observation period (in | Calculated by the following equation: [End Date] - [Start Date] + 1. |
| days) | |
| Treatment duration (in | A total of ([End Date] - [Start Date] + 1) in the number of actual administration |
| days) | days, excluding washout period. |
| Mean daily dose | Calculated by the following equation: Total of ([Daily Dose] × [Total Period of |
| | Treatment with the Dose]) / [Observation Period]. See the above for calculation |
| | of observation period. |
| Concomitant medication | A drug used during the surveillance period. However, concomitant medications |

| Item | Definition |
|---|---|
| | exclude drugs used for adverse events occurring during the period. |
| Antihyperlipidemic drug | A drug starting with any of the following drug codes: 218, 2190006, 2190101, |
| | 2190102, 2190103, 2190104, 290006, 3133001, 3133400, 3399004. |
| Statins drug | A drug starting with any of the following drug codes: 2189010, 2189011, |
| | 2189012, 2189015, 2189016, 2189017. |
| Fibrate drug | A drug starting with drug code: 2183. |
| Intestinal transporter | A drug starting with drug code: 2189018. |
| inhibitor | |
| Anion-exchange resin | A drug starting with any of the following drug codes: 2189009, 2189014. |
| Nicotinic acid derivative | A drug starting with any of the following drug codes: 2189004, 2189005, |
| | 2190006. |
| Probucol | A drug starting with drug code: 2189008. |
| Ethyl icosapentate (EPA) | A drug starting with drug code: 3399004. |
| Cardiovascular drug | A drug starting with drug code: 21. |
| Antidiabetic drug | A drug starting with any of the following drug codes: 396, 2492, 249941. |
| Anticoagulant drug | A drug starting with any of the following drug codes: 333, 2190408, 6343424. |
| Antiplatelet drug | A drug starting with any of the following drug codes: 3399 (excluding |
| | 3399004), 2171010, 2171402. |
| LDL cholesterol | Calculated the equation below if the patient is fasting at the time of blood |
| (Friedewald formula) | collection for laboratory testing with triglyceride 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol - triglyceride / 5 |
| Non-HDL cholesterol | Calculated by the equation below if triglyceride is 400 mg/dL or over. Indicated |
| (mg/dL) | by rounding off to an integer alone. |
| | Total cholesterol - HDL cholesterol |
| TC/LDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | Total cholesterol / LDL cholesterol (Friedewald formula) |
| LDL-C/HDL-C ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / HDL cholesterol |
| LDL-C/Apo-B ratio | Calculated by the equation below. Indicated by rounding off to the first decimal |
| | place. |
| | LDL cholesterol (Friedewald formula) / Apo-B |
| Summary statistics | Mean value, standard deviation, minimum value, first quartile, median, third |
| | quartile, maximum value |

#### 1.2 Number of Display Digits

| Item | Definition |
|---|---|
| Percentage (%) | Rate of patients with ADRs: |
| | Indicated by rounding off to the second decimal place. |
| | Other than above: |
| | Indicated by rounding off to the first decimal place. |
| Summary statistics | Mean value: |
| (Mean value/standard | Indicated by rounding off to the first digit below the raw numerical data. |
| deviation) | Standard deviation: |
| | Indicated by rounding off to the second digit below the raw numerical data. |
| p value | Indicated by rounding down to the third decimal place. |
| | Expressed as p<0.001 when rounding down at the forth decimal place makes the |
| | figure below 0.001. |

#### 1.3 Level of Significance

Two-sided 5%

#### 1.4 Handling of Evaluation Timepoint Data

The evaluation timepoints are the start of treatment with the Drug (baseline), Month 3, Month 6, Month 9, Month 12, and final evaluation timepoint.

If multiple data exist within each evaluation timepoint, calculate absolute values of difference in measurement intervals from the basic day count and adopt the minimum absolute value as date for that evaluation timepoint. If all the absolute values are the same, adopt one for the latest date of measurement. Measurements should not be adopted that have been obtained after completion of treatment with the Drug. The final evaluation timepoint measurement should be one taken on the latest date within 405 days elapsed since the start date (including values measured during washout period). Note that the number days elapsed since the start date should be counted with the start date as day 0 and the previous day as day -1.

| Evaluation Timepoint | Tolerance<br>(Number of Days Since Baseline) | Basic Day Count |
|---|---|---|
| Baseline | -90 to 0 | 0 |
| Month 3 | 1 to 135 | 90 |
| Month 6 | 136 to 225 | 180 |
| Month 9 | 226 to 315 | 270 |
| Month 12 | 316 to 405 | 360 |
| Final evaluation | 1 to 405 | - |
| timepoint | | |

#### 2.0 Results of Special Drug Use Surveillance (Survey 1)

<Lotriga Granular Capsules Special Drug Use Surveillance [long-term use survey]>

#### 2.1 Patient Breakdown (Patient Disposition)

| Statistical Analysis | Enrolled patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Number of enrolled patients, number of patient enrollment sites, number of patients |
| Statistical Analysis | with eCRFs collected, number of patients with eCRFs uncollected, number of locked |
| | patients, number of unlocked patients, number of safety-evaluable patients, number of |
| | safety-unevaluable patients, number of efficacy-evaluable patients, number of |
| | efficacy-unevaluable patients |
| | Do not double-count the same medical institution with different participating clinical |
| | departments when counting the number of patient enrollment sites. |
| | Count the number of patients per reason for not collecting and total the numbers when |
| | the number of patients with eCRFs uncollected. |
| | Count the number of patients per reason for exclusion and total the numbers when |
| | counting the numbers of safety- and efficacy-unevaluable patients. |
| Figure/Table No. | Figure 2.1, Table 2.1 |

#### 2.2 Patient Demographics

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |

Details of Statistical Analysis Categorize the patient population by the following categories for each item and compile the number of patients and incidence.

| Item Name | Category |
|---|---|
| Sex | Male, Female |
| Age | Summary statistics |
| | Minimum age to 64 years, 65 to 74 years, 75 years to |
| | maximum age, Unknown |
| Treatment category | Outpatient, inpatient |
| Weight | Summary statistics |
| | Less than 40 kg, 40 to less than 50 kg, 50 to less than |
| | 60 kg, 60 to less than 70 kg, 70 to less than 80 kg, 80 |
| | to less than 90 kg, 90 kg or over, Not measured |
| BMI | Summary statistics |
| | Less than $18.5 \text{ kg/m}^2$ , $18.5 \text{ to less than } 25 \text{ kg/m}^2$ , $25 \text{ to}$ |
| | less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| Complications | No, Yes |
| | Hypertension, Diabetic, Liver disorder, Kidney |
| | disorder, Cardiac disorders [myocardial infarction, |
| Complication | angina pectoris, atrial fibrillation, others], |
| breakdown | Cerebrovascular diseases [hemorrhagic |
| | cerebrovascular disease, ischemic cerebrovascular |
| | disease, others], Bleeding-related event, Others |
| Drinking history | |
| (Does the patient | |
| drink alcoholic | Yes, No, Unknown |
| beverages nearly | |
| every day?) | |
| | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | to less than 500 mg/dL, 500mg/dL or over, Not |
| F (: (:1 :1 :1 ) | measured |
| Fasting triglyceride at baseline (mg/dL) | |
| | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 |
| | to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | 750 mg/dL or over, Not measured |

| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured |
|---|---|---|
| | | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Smoking history | Never, Current, Former, Unknown |
| | Menopausal status (only for female) | No, Yes |
| | Hypersensitivity disposition | No, Yes, Unknown |
| | Disease duration | Summary statistics |
| | | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence<br>of surgery within one<br>month before baseline | No, Yes |
| | Pregnancy status<br>during treatment (only<br>for female) | No, Yes |
| Figure/Table No. Table 2.2 | | |
#### 2.3 Treatment Details

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize the patient population by the following categories for each item and | |
| Statistical Analysis | compile the number of patients and incidence. | |
| | Item Name | Category |
| | Initial dose | 2 g, 4 g, Other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant | |
| | medications (during | No, Yes |
| | observation period) | |
| | Breakdown of concomitant medications (during | Antihyperlipidemic drugs [statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others], Cardiovascular drugs, Antidiabetic |
| | observation period) | drugs, Anticoagulant/antiplatelet drugs [anticoagulant drugs, antiplatelet drugs] |
| | Completion of treatment with the Drug | No, Yes, Unknown |
| | Reason for treatment | Treatment goal achieved, AE developing, Patient no |
| | completion | longer visiting hospital due to hospital transfer or |
| | | otherwise, Insufficient effect, Other |
| Figure/Table No. | Table 2.3 | |

# 2.4 Safety Statistical Analysis

# 2.4.1 Onset Status of Adverse Drug Reactions or Infections (Exhibit 2)

| | 1 | |
|---|---|---|
| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in | |
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the | |
| | Adverse Drug Reactions section of the package insert) and this special drug use | |
| | surveillance | |
| Details of | Compile the following items for the prior-approval status and per survey unit period | |
| Statistical Analysis | of the special drug use surveil | llance. |
| | | r of study sites,' 'number of surveyed patients,' 'number |
| | | number of ADRs' should cover safety-evaluable patients |
| | locked during each survey un | • |
| | Item Name | Details of Statistical Analysis |
| | Item Name | Number of medical institutions that have collected |
| | Number of study sites | eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients with ADRs | Number of patients in which ADRs occurred. |
| | Number of ADRs | Number of ADRs that occurred. Every PT occurring should be counted as one event. |
| | Rate of patients with ADRs | Described in section 1.1. |
| | ADR type | Categorize by SOC and compile ADRs by PT in each category. In the case of laboratory testing, categorize by SOC, summarize by HLGT, and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. At PT level, the numbers of ADRs should be presented by PT code in ascending order. If adverse drug reactions (LLTs) under the same PT occur more than once in the same patient, they should be counted as one PT. |
| | Cumulative total for special drug use surveillance | A respective total of the numbers of study sites and patients per survey unit period. Do not double-count the same medical institution when counting the number of study sites. A combination of the total for the prior-approval status and the cumulative total for the special drug |
| | Combined total | use surveillance. Do not double-count the same medical institution when counting the number of study sites. |
| Figure/Table No. | Table 2.4.1 | |

# 2.4.2 Onset Status of Adverse Drug Reactions/Infections in Safety-Unevaluable Patients (Exhibit 2)

| Statistical Analysis | Safety-unevaluable patients in clinical studies before approval (total of patients in | |
|---|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the | |
| | Adverse Drug Reactions section of the package insert) and this specified drug use | |
| | surveillance | |
| Details of | Compile the following items. | |
| Statistical Analysis | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-unevaluable patients. |
| | Number of patients with ADRs | Number of patients in which ADRs occurred. |
| | Number of ADRs | Number of ADRs that have occurred. Every PT occurring should be counted as one event. |
| | Rate of patients with ADRs | Described in section 1.1. |
| | ADR type | Categorize by SOC and compile ADRs by PT in each category. In the case of laboratory testing, categorize by SOC, summarize by HLGT, and compile ADRs by PT. At SOC level, the numbers and rates of patients with ADRs should be presented by SOC internationally agreed order. At PT level, the numbers of ADRs should be presented by PT code in ascending order. If adverse drug reactions (LLTs) under the same PT occur more than once in the same patient, they should be counted as one PT. |
| | Combined total | A combination of the totals for the prior-approval status and for the special drug use surveillance. Do not double-count the same medical institution when counting the number of study sites. |
| Figure/Table No. | Table 2.4.2 | |

#### 2.4.3 Onset Status of AE

| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in |
|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the |
| | Adverse Drug Reactions section of the package insert) and this special drug use |
| | surveillance |
| Details of | The compilation method is the same as described in section 2.4.1. However, adverse |
| Statistical Analysis | drug reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.3 |

# 2.4.4 Onset Status of Adverse Events in Safety-Unevaluable Patients

| Statistical Analysis | Safety-unevaluable patients in clinical studies before approval (total of patients in |
|---|---|
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the |
| | Adverse Drug Reactions section of the package insert) and this specified drug use |
| | surveillance |
| Details of | Compilation method is the same as described in section 2.4.2. However, adverse drug |
| Statistical Analysis | reactions should be replaced by adverse events. |
| Figure/Table No. | Table 2.4.4 |

# 2.4.5 Onset Status of Adverse Drug Reactions or Infections by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADRs by the following categories for each item and compile ADR types. | |
| Statistical Analysis | Item Name Details of Statistical Analysis | |
| | Number of patients Compile the number of patients with ADRs. | |
| | Number of ADRs At SOC, the number of ADRs should be compiled by totaling associated PTs that occurred. At PT level, every PT occurring should be counted as one event. | |
| | Item Name Category | |
| | Seriousness Serious, Not serious, N/A | |
| | Onset time 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over, Unknown | О |
| | Outcome Resolved, Resolved, Resolved with sequelaed Death, Unknown | е, |
| Figure/Table No. | Table 2.4.5 | |

# 2.4.6 Onset Status of Adverse Events by Seriousness, Onset Time, and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize AEs | by the following categories for each item and compile AE types. |
| Statistical Analysis | The compilation | n method of ADR types is the same as described in section 2.4.5. |
| | However, adver | rse drug reactions should be replaced by adverse events. |
| | Item Name | Category |
| | Seriousness | Serious, Not serious, N/A |
| | On set time | 1 to 15 days, 16 to 30 days, 31 to 90 days, 91 to 180 days, 181 to |
| | Onset time | 360 days, 361 days or over, Unknown |
| | Outcome | Resolved, Resolving, Not resolved, Resolved with sequelae, |
| | Outcome | Death, Unknown |
| | Causal | Related, Not related, Unevaluable |
| | | If adverse drug reactions (LLTs) occur more than once in the same |
| | relationship with the Drug | patient, they should be counted as one event in the following |
| | | order of priority: |
| | | (1) Related, (2) Unevaluable, (3) Not related |
| Figure/Table No. | Table 2.4.6 | |

# 2.4.7 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Seriousness, Onset Time,

#### and Outcome

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Categorize adverse drug reactions (bleeding-related events) by the following |
| Statistical Analysis | categories for each item, and count the types of adverse drug reactions |
| | (bleeding-related events). |
| | The categories and the compilation method of adverse drug reactions are the same as |
| | described in section 2.4.5. |
| Figure/Table No. | Table 2.4.7 |

# 2.4.8 Rate of Patients of Adverse Drug Reactions or Infections by Factor of Patient Demographics and Treatment Details

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance | |
|---|---|---|
| Set | | |
| Details of | Categorize ADRs by the following categories for each item and compile the rate of | |
| Statistical Analysis | patients with ADRs (point estimate and 95% confidence interval). | |
| | Perform Fisher's exact test for items having categories without rank order, and | |
| | Mann-Whitney U test for | items having categories with rank order. |
| | Item Name | Category |
| | Sex | Male, Female |
| | A 92 | Minimum age to 64 years, 65 to 74 years, 75 years to |
| | Age | maximum age, Unknown |
| | | Less than 40 kg, 40 to less than 50 kg, 50 to less than |
| | Weight | 60 kg, 60 to less than 70 kg, 70 to less than 80 kg, 80 |
| | | to less than 90 kg, 90 kg or over, not measured |
| | DIG | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to |
| | BMI | less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Complications | No, Yes |
| | | Hypertension, Diabetic, Liver disorder, Kidney |
| | | disorder, Cardiac disorders [myocardial infarction, |
| | Complication | angina pectoris, atrial fibrillation, others], |
| | breakdown | Cerebrovascular diseases [hemorrhagic |
| | | cerebrovascular disease, ischaemic cerebrovascular |
| | | disease, others], Bleeding-related event, Others |
| | Drinking history | 7 |
| | (Does the patien | |
| | drink alcoholic | Yes, No, Unknown |
| | beverages nearly | , |
| | every day?) | |
| | | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 |
| | | to less than 500 mg/dL, 500mg/dL or over, Not |
| | Fasting triglyceride a | |
| | baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 |
| | | to less than 500 mg/dL, 500 to less than 750 mg/dL, |
| | | 750 mg/dL or over, Not measured |

| | Item Name | Category |
|---|---|---|
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500mg/dL or over, Not measured |
| | | Less than 150 mg/dL, 150 to less than 400mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over, Not measured |
| | Smoking history | Never, Current, Former, Unknown |
| | Menopausal status (only for female) | No, Yes |
| | Hypersensitivity disposition | No, Yes, Unknown |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Presence or absence of surgery within one month before baseline | No, Yes |
| | Pregnancy status during treatment (only for female) | No, Yes |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) | No, Yes |
| | Breakdown of concomitant medications (during observation period) | Antihyperlipidemic drugs [statins drugs, fibrate drugs, intestinal transporter inhibitors, anion-exchange resin, nicotinic acid derivatives, probucol, ethyl icosapentate (EPA), others], Cardiovascular drugs, Antidiabetic drugs, Anticoagulant/antiplatelet drugs [anticoagulant drugs, antiplatelet drugs] |
| Figure/Table No. | Table 2.4.8 | |

#### 2.4.9 Onset Status of Adverse Drug Reactions or Infections by Age Group

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Classify the patient population into 64 years or below, 65 to 74 years, and 75 years or |
| Statistical Analysis | over, and compile ADR types. |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.9 |

# 2.4.10 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Liver

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of liver complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.10 |

# 2.4.11 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Kidney

#### Complications

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of kidney complications. |
| Statistical Analysis | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.11 |

# 2.4.12 Onset Status of Adverse Drug Reactions or Infections by Presence or Absence of Concomitant

#### Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile ADR types by presence or absence of concomitant anticoagulant and/or |
| Statistical Analysis | antiplatelet drugs (Both, Anticoagulant only, Antiplatelet only, Neither). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.12 |

# 2.4.13 Onset Status of Adverse Drug Reactions (Bleeding-Related Events) by Presence or Absence of Concomitant Anticoagulant and/or Antiplatelet Drugs

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Compile the types of adverse drug reactions (bleeding-related events) by presence or |
| Statistical Analysis | absence of concomitant anticoagulant and/or antiplatelet drugs (Both, Anticoagulant |
| | only, Antiplatelet only, Neither). |
| | The compilation method of the types of adverse drug reactions is the same as |
| | described in section 2.4.1. |
| Figure/Table No. | Table 2.4.13 |

# 2.4.14 Onset Status of Adverse Drug Reactions or Infections by Baseline Fasting Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose fasting |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline fasting triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.14 |

#### 2.4.15 Onset Status of Adverse Drug Reactions or Infections by Baseline Random Triglyceride Level

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance whose random |
|---|---|
| Set | triglyceride levels were measured at baseline |
| Details of | Compile ADR types by baseline random triglyceride level (Less than 150 mg/dL, 150 |
| Statistical Analysis | to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 |
| | mg/dL or over). |
| | The compilation method of ADR types is the same as described in section 2.4.1. |
| Figure/Table No. | Table 2.4.15 |

#### 2.4.16 Changes in Laboratory Test Values (Glucose Metabolism)

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseli |
| | In addition, calculate the 95% confidence interval for the mean value for variation |
| | from baseline. Also perform the corresponding t-test. |
| Figure/Table No. | Table 2.4.16 |

# 2.4.17 Changes in Laboratory Test Values (Glucose Metabolism) < With Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variations |
| | from baseline. Also perform the corresponding t-test. |
| Remarks | Stratification factor: With diabetic complications |
| Figure/Table No. | Table 2.4.17 |

# 2.4.18 Changes in Laboratory Test Values (Glucose Metabolism) < Without Diabetic Complications>

| Statistical Analysis | Safety-evaluable patients in this special drug use surveillance |
|---|---|
| Set | |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting blood glucose |
| Statistical Analysis | (mg/dL) and HbA1c (NGSP value) (%) measurements and variations from baseline. |
| | In addition, calculate the 95% confidence interval for the mean value for variation |
| | from baseline. Also perform the corresponding t-test. |
| Remarks | Stratification factor: Without diabetic complications |
| Figure/Table No. | Table 2.4.18 |

# 2.5 Efficacy Statistical Analysis

# 2.5.1 Changes in Laboratory Test Values (Fasting Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for fasting measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), total cholesterol |
| | (mg/dL), LDL cholesterol (direct measurement) (mg/dL), LDL cholesterol |
| | (Friedewald formula) (mg/dL), HDL cholesterol (mg/dL), non-HDL cholesterol |
| | (mg/dL), VLDL cholesterol (mg/dL), Apo-AI (mg/dL), Apo-B (mg/dL), Apo-CIII |
| | (mg/dL), lipoprotein(a) (mg/dL), and remnant lipoprotein cholesterol (mg/dL). In |
| | addition, calculate the 95% confidence interval for the mean value for rates of change |
| | from baseline (%). Also perform the corresponding t-test. |
| Figure/Table No. | Table 2.5.1 |

# 2.5.2 Changes in Laboratory Test Values (Random Lipid)

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom random |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for random measurements |
| Statistical Analysis | and rates of change from baseline (%) of triglyceride (mg/dL), total cholesterol |
| | (mg/dL), LDL cholesterol (direct measurement) (mg/dL), HDL cholesterol (mg/dL), |
| | $non\text{-}HDL\ cholesterol\ (mg/dL),\ VLDL\ cholesterol,\ Apo\text{-}AI\ (mg/dL),\ Apo\text{-}B\ (mg/dL),$ |
| | Apo-CIII (mg/dL), lipoprotein(a) (mg/dL), and remnant lipoprotein cholesterol |
| | (mg/dL). In addition, calculate the 95% confidence interval for the mean value for |
| | rates of change from baseline (%). Also perform the corresponding t-test. |
| Figure/Table No. | Table 2.5.2 |

# 2.5.3 Changes in Fasting Lipid-Related Ratio

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting |
|---|---|
| Set | blood collection was performed at baseline |
| Details of | Calculate summary statistics at each evaluation timepoint for TC/LDL-C, |
| Statistical Analysis | LDL-C/HDL-C, and LDL-C/Apo-B. |
| Figure/Table No. | Table 2.5.3 |

# 2.5.4 Changes in Fasting Triglyceride by Factor of Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom fasting | |
|---|---|---|
| Set | blood collection was performed at baseline | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of fasting | |
| | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age | Minimum age to 64 years, 65 to 74 years, 75 years to maximum age, Unknown |
| | Weight | Less than 40 kg, 40 to less than 50 kg, 50 to less than 60 kg, 60 to less than 70 kg, 70 to less than 80 kg, 80 to less than 90 kg, 90 kg or over, not measured |
| | BMI | Less than 18.5kg/m <sup>2</sup> , 18.5 to less than 25kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Fasting triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over |
| | Menopausal status (only for female) | No, Yes |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) (antihyperlipidemic drugs) | No, Yes |
| | Breakdown of concomitant medications (during observation period) (antihyperlipidemic drugs) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |
| Figure/Table No. | Table 2.5.4 | |

# 2.5.5 Changes in Random Triglyceride by Factor of Patient Demographics and Treatment Details

| Statistical Analysis | Efficacy-evaluable patients in this special drug use surveillance for whom random | |
|---|---|---|
| Set | blood collection was performed at baseline | |
| Details of | Calculate summary statistics by stratification for each item for baseline and final | |
| Statistical Analysis | evaluation timepoint measurements and rates of change from baseline (%) of random | |
| J | triglyceride. | |
| | Item Name | Category |
| | Sex | Male, Female |
| | Age<br>Weight | Minimum age to 64 years, 65 to 74 years, 75 years to |
| | | maximum age, Unknown |
| | | Less than 40 kg, 40 to less than 50 kg, 50 to less than |
| | | 60 kg, 60 to less than 70 kg, 70 to less than 80 kg, 80 |
| | | to less than 90 kg, 90 kg or over, not measured |
| | BMI | Less than 18.5 kg/m <sup>2</sup> , 18.5 to less than 25 kg/m <sup>2</sup> , 25 to less than 30 kg/m <sup>2</sup> , 30 kg/m <sup>2</sup> or over, unknown |
| | Random triglyceride at baseline (mg/dL) | Less than 150 mg/dL, 150 to less than 400 mg/dL, 400 to less than 500 mg/dL, 500 to less than 750 mg/dL, 750 mg/dL or over |
| | Menopausal status (only for female) | No, Yes |
| | Disease duration | Less than 1 year, 1 to less than 3 years, 3 to less than 5 years, 5 years or over, Unknown |
| | Initial dose | 2 g, 4 g, other |
| | Change in daily dose | No, Yes |
| | Breakdown of change in daily dose | $2 \text{ g} \rightarrow 4 \text{ g}, 4 \text{ g} \rightarrow 2 \text{ g}, \text{Other}$ |
| | Mean daily dose | Less than 2 g, 2 to less than 4 g, 4 to less than 6 g, 6 g or over |
| | Treatment duration | 1 to 30 days, 31 to 90 days, 91 to 180 days, 181 to 360 days, 361 days or over |
| | Concomitant medications (during observation period) (antihyperlipidemic drugs) | No, Yes |
| | Breakdown of concomitant medications (during observation period) (antihyperlipidemic drugs) | Statins drugs, Fibrate drugs, Intestinal transporter inhibitors, Anion-exchange resin, Nicotinic acid derivatives, Probucol, Ethyl icosapentate (EPA), Others |
| Figure/Table No. | Table 2.5.5 | <u>, </u> |

# 3.0 Summary of Onset Status of Serious Adverse Events (Exhibit 2-2)

| Summary of Ons | et Status of Serious Advers | e Events (Exhibit 2-2) |
|---|---|---|
| Statistical Analysis | Safety-evaluable patients in clinical studies before approval (total of patients in | |
| Set | clinical studies inside and outside Japan used for safety evaluation stated in the | |
| Set | Adverse Drug Reactions section of the package insert) and this special drug use | |
| | surveillance | seemen of the property and the special and the |
| Details of | | ns per survey unit period of the prior-approval status and of |
| Statistical Analysis | the use-results surveillance/special drug use surveillance. | |
| | Statistical analysis of 'number of study sites,' 'number of surveyed patients,' 'number | |
| | of patients with AEs,' and 'number of AEs' should cover safety-evaluable patients | |
| | locked during each survey | |
| | Item Name | Details of Statistical Analysis |
| | Number of study sites | Number of medical institutions that have collected eCRFs |
| | Number of surveyed patients | Number of safety-evaluable patients. |
| | Number of patients | Number of patients with SAEs |
| | Number of SAEs | Number of SAEs |
| | | Every PT occurring should be counted as one event. |
| | | Calculated by the following equation: [Number of |
| | Rate of patients | Patients with SAEs] / [Number of Safety-Evaluable |
| | | Patients] × 100. |
| | SAE type | Categorize by SOC and compile ADRs by PT in each category. In the case of laboratory testing, categorize by SOC, summarize by HLGT, and compile ADRs by PT. At SOC level, the numbers and rates of patients with AEs should be presented by SOC internationally agreed order. At PT level, the numbers of ADRs should be presented by PT code in ascending order. If adverse drug reactions (LLTs) under the same PT occur more than once in the same patient, they should be counted as one PT. The number of SAEs of which causal relationship to the Drug has been denied should be entered in the [ ] brackets. |
| | Cumulative total Combined total | A respective total of the numbers of study sites and patients per survey unit period. Do not double-count the same medical institution when counting the number of study sites. A combination of the total for the prior-approval status and the cumulative total. Do not double-count the same medical institution |
| | | when counting the number of study sites. |
| Figure/Table No. | Table 3.0 | |